

# Statistical Analysis Plan

## **ABX464-301**

# Phase IIa study of ABX464 in moderate to severe active Rheumatoid Arthritis patients

Prepared for:

## **ABIVAX**

5 rue de la Baume

75008 Paris - France

Tel: +33 (0) I 53 83 08 41

Fax: +33 (0) I 53 83 07 48

Prepared by:

## **ORION Clinical**

7 Bath Road, Slough

Berkshire SLI 3UE UK

Tel: +44 (0) 1753 578080

Fax: +44 (0) 1753 578081

CONFIDENTIAL

Version Author

Final 1.0 Lilla Hanák



# Statistical Analysis Plan

## ABX464-301

# Phase IIa study of ABX464 in moderate to severe active Rheumatoid Arthritis patients

| Author: | Lilla Hanák | |
|---|---|---|
| Version: | Final 1.0 | |
| The undersi<br>requirement | gned have reviewed and revised this SAP and find it to be one constant. | consistent with the study |
| Paul Gines | te, Vice President, Clinical Operations, Abivax | Date |
| Lilla Hanál | ς, Statistician, Simbec-Orion Group Ltd | Date |
| | , | |
| Virginie C | ombe, Head of Statistics, Simbec-Orion Group Ltd | Date |



# **TABLE OF CONTENTS**

| 1 | INTRO | DUCTION | 8 |
|---|---|---|---|
| | 1.1 | General | 8 |
| | 1.2 | Changes from Protocol | 8 |
| | 1.3 | Changes from Previous Versions of the SAP | 8 |
| 2 | STUDY | OBJECTIVES | 8 |
| | 2.1 | Primary Objective | 8 |
| | 2.2 | Secondary Objectives | 8 |
| 3 | STUDY | DESIGN | 9 |
| | 3.1 | Overview | 9 |
| | 3.2 | Inclusion and Exclusion Criteria | 10 |
| | 3.2.1 | Inclusion criteria | 10 |
| | 3.2.2 | Exclusion criteria | 11 |
| | 3.3 | Study Treatment | 13 |
| | 3.4 | Study Timepoints | 13 |
| | 3.5 | Sample Size Considerations | 14 |
| | 3.6 | Randomisation | 15 |
| 4 | STUDY | VARIABLES AND COVARIATES | 15 |
| | 4.1 | Primary Variable | 15 |
| | 4.2 | Secondary Efficacy Variables | 15 |
| | 4.2.1 | Main Secondary Efficacy Endpoint | 15 |
| | 4.2.2 | Other secondary endpoints | 16 |
| | 4.3 | Pharmacokinetic Variables | 17 |
| | 4.4 | Pharmacodynamic Variables | 17 |
| | 4.5 | Other Outcome Variables | 17 |
| | 4.6 | Safety Variables | 17 |
| 5 | DEFINI | TIONS AND DERIVED VARIABLES | 17 |
| | 5.1 | Definitions | 17 |
| | 5.2 | Derived variables | 18 |
| | 5.2.1 | Disease Activity Score (DAS) 28-CRP (DAS28-CRP) and DAS28-ESR | 18 |
| | 5.2.2 | Simplified Disease Activity Index (SDAI) | 18 |



# GROUP

| | 5.2.3 | Clinical Disease Activity Index (CDAI) | 18 |
|---|---|---|---|
| | 5.2.4 | Categorical DAS28-CRP response | 19 |
| | 5.2.5 | DAS28-ESR remission | 19 |
| | 5.2.6 | Low Disease Activity (LDA) | 19 |
| | 5.2.7 | SDAI remission | 19 |
| | 5.2.8 | CDAI remission | 19 |
| | 5.2.9 | ACR/EULAR remission: | 19 |
| | 5.2.10 | Categorical ACR20/50/70 response | 19 |
| | 5.2.11 | Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue: | 21 |
| 6 | ANALYS | SIS SETS | 22 |
| | 6. l | Full Analysis Set | 22 |
| | 6.2 | Safety Set | 22 |
| | 6.3 | Efficacy Set | 22 |
| | 6.3.1 | "raw" Efficacy Set | 22 |
| | 6.3.2 | Efficacy Set with imputation | 22 |
| | 6.4 | Per Protocol Set | 22 |
| 7 | SAFETY | MONITORING | 23 |
| 8 | INTERIN | ∕I ANALYSES | 24 |
| 9 | DATA | | 24 |
| | 9.1 | eCRF Data | 24 |
| | 9.2 | External Data | 24 |
| | 9.2.1 | Laboratory Data | 24 |
| | 9.2.2 | Other non-CRF data | 25 |
| | 9.3 | Randomisation list | 25 |
| | 9.4 | Programming and Data Review | 26 |
| 10 | STATIST | FICAL METHODS | 26 |
| | 10.1 | General Principles | 26 |
| | 10.2 | Stratification and Covariate Adjustment | 28 |
| | 10.3 | Interactions | 28 |
| | 10.4 | Missing Data | 28 |
| | 10.5 | Pooling of Sites | 28 |
| | 10.6 | Multiple Comparisons | 28 |
| | 10.7 | Subgroup Analyses | 28 |
| | 10.8 | Statistical Issues | 28 |
| 11 | STATIST | TICAL OUTPUT | 29 |



# GROUP

| | 11.1 | Patient Disposition | 29 |
|----|---------|------------------------------------------------|-----|
| | 11.2 | Patient Characteristics at Baseline | 29 |
| | 11.2.1 | Demographic and Baseline Characteristics | 29 |
| | 11.2.2 | Medical History and Current Medical Conditions | 29 |
| | 11.3 | Efficacy Analyses | 29 |
| | 11.3.1 | Primary Variable | 30 |
| | 11.3.2 | Secondary Variables | 30 |
| | 11.4 | PK Analyses | 31 |
| | 11.5 | PD analyses | 31 |
| | 11.6 | Safety Analyses | 31 |
| | 11.6.1 | Adverse Events | 31 |
| | 11.6.2 | Laboratory Data | 33 |
| | 11.6.3 | Vital Signs | 33 |
| | 11.6.4 | Physical Examination | 34 |
| | 11.6.5 | Electrocardiogram | 34 |
| | 11.7 | Study Drug Exposure and Compliance | 34 |
| | 11.8 | Prior and Concomitant Medication | 34 |
| 12 | VALIDA | TION | 36 |
| 13 | LITERAT | URE CITATIONS/REFERENCES | 36 |
| 14 | LIST OF | TABLES, FIGURES AND LISTINGS | 37 |
| | 14.1 | List of Tables | 37 |
| | 14.2 | List of Listings | 39 |
| 15 | SHELLS | FOR TABLES, FIGURES AND LISTINGS | 40 |
| 16 | APPEND | DICES | 101 |
| | 16.1 | Study flowchart | 101 |



# **GLOSSARY OF ABBREVIATIONS**

| %CV | Coefficient of Variation |
|--------|------------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine Transaminase (also SGPT) |
| AM | Arithmetic Mean |
| ANCOVA | Analysis of Covariance |
| ANOVA | Analysis of Variance |
| AST | Aspartate Transaminase (also SGOT) |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CR | Complete Response |
| CRF | Case Report Form |
| CRO | Clinical Research Organisation |
| CS | Clinically Significant |
| CSR | Clinical Study Report |
| CTCAE | Common Toxicity Criteria Adverse Event |
| CV | Coefficient of Variation |
| DMP | Data Management Plan |
| DOB | Date of Birth |
| DRM | Data Review Meeting |
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| GM | Geometric Mean |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IMP | Investigational Medicinal Product |
| IQR | Interquartile Range |
| ITT | Intention-to-treat |



| IV | Intravenous |
|---------|----------------------------------------------|
| LambdaZ | Terminal phase rate constant |
| LOCF | Last Observation Carried Forward |
| LS Mean | Least Squares Mean |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| ml | Millilitre |
| N | Number of Patients |
| n | Number of Events |
| NCS | Not clinically significant |
| od | Once daily |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PP | Per Protocol |
| PR | Partial Response |
| PT | Preferred Term |
| q12h | Every 12 hours |
| QC | Quality Control |
| QoL | Quality of Life |
| RA | Accumulation ratio |
| RBC | Red Blood Cell |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| VAS | Visual Analogue Scale |
| WBC | White Blood Cell |
| μg | Microgram |
| TEAE | Treatment Emergent Adverse Event |
| VAS | Visual Analogue Scale |



## 1 INTRODUCTION

#### 1.1 GENERAL

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under ABIVAX Protocol ABX464-301 and should be read in conjunction with the study protocol and case report form (CRF).

This version of the plan has been developed using the protocol Version 4.0 dated 24OCT2019 (and CRF/ Electronic Data Capture (EDC) specifications dated 06FEB2020. Any further changes to the protocol or CRF will be reviewed for potential impact on the SAP which will be amended if it is deemed necessary.

At the time of writing this version of the SAP, recruitment is ongoing.

Draft I was reviewed by the Orion project manager, medical writer and statistical reviewer. The analysis plan will be finalised and approved by the sponsor prior to unblinding of study treatment codes for the planned interim analysis and prior to database lock.

#### 1.2 CHANGES FROM PROTOCOL

It is stated in the protocol that "Analysis of efficacy data will be carried out in the Full Analysis Set in which subjects who prematurely terminate the study will be considered failures."

Sponsor requested by email having 2 efficacy set.

## 1.3 CHANGES FROM PREVIOUS VERSIONS OF THE SAP

No previous versions of the SAP exist.

## 2 STUDY OBJECTIVES

#### 2.1 PRIMARY OBJECTIVE

The primary objective of the study is to evaluate the safety of ABX464 given at two different doses (100mg and 50 mg) vs placebo in combination with MTX when administered once daily in patients with moderate to severe active Rheumatoid Arthritis.

#### 2.2 SECONDARY OBJECTIVES

The secondary objectives are the followings:



- To evaluate the effects of the different dose groups of ABX464 at Week 2, Week 4, Week 8
  and Week 12 on the American College of Rheumatology (ACR) 20/50/70 response and each of
  its components versus placebo;
- To evaluate the effects of the different dose groups of ABX464 at Week 2, Week 4, Week 8
  and Week 12 on disease activity scores (DAS28 scores, simplified disease activity score [SDAI]
  and clinical disease activity score [CDAI]) versus placebo;
- To evaluate the effects of the different dose groups of ABX464 at Week 2, Week 4, Week 8 and Week 12 on clinical response (DAS28 EULAR good and moderate responses), Low Disease Activity (LDA) or remission (DAS28-ESR remission, ACR/EULAR remission, SDAI and CDAI remission) versus placebo;
- To evaluate the effects of the different dose groups of ABX464 at Week 2, Week 4, Week 8
   and Week 12 on the Patient Reported Outcome (PRO), Healthy Assessment Questionnaire –
   Disability Index (HAQ-DI);
- To evaluate the expression of miR-124 in total blood (determined by qPCR) at baseline and Week 8;
- To evaluate the effects of different dose groups of ABX464 at Week 8 on miR-124 expression in total blood versus placebo;
- To assess the pharmacokinetics of the ABX464 and its main active metabolite N-Glu-ABX464 after oral administration of different daily doses of ABX464 in patients with Rheumatoid Arthritis.

## 3 STUDY DESIGN

## 3.1 OVERVIEW

This Phase IIa study is a randomized, double blind, placebo controlled, parallel group, multiple dose study on ABX464 in combination with methotrexate (MTX), in patients with moderate to severe active Rheumatoid Arthritis who have inadequate response to MTX or/and to an anti- tumor necrosis factor alpha (TNF $\alpha$ ) therapy, or intolerance to anti-TNF $\alpha$  therapy.

Several experimental and clinical endpoints will be assessed to obtain information on preliminary efficacy in patients with moderate to severe active Rheumatoid Arthritis. Although no formal hypothesis will be tested, these endpoints will enable a broader understanding of the mechanism of action and potential for clinical efficacy of ABX464 in Rheumatoid Arthritis. No interim analysis is planned.

Up to 60 patients will be randomized in this study. These patients will be enrolled in approximately 20 sites located in Europe. At the beginning, the first 6 patients will be randomized to receive either ABX464 50mg (n=4) or its matching placebo (n=2). The Data Safety Monitoring Board (DSMB) will review the safety of these first 6 patients dosed for at least 2 weeks. Once the DSMB recommendation is granted, the next patients will be randomized to receive either ABX464 50mg, ABX464 100mg or placebo. Then, a second DSMB meeting will be held after the next 6 patients are randomized to check the tolerability



of the 100mg dose. Once the DSMB recommendation is granted, the next patients will be randomized to receive either ABX464 50mg, ABX464 100mg or placebo. The study randomization ratio is 1:1:1.

The recruitment period is between Q2 2019 and Q3 2020, the overall study period is between Q2 2019 and Q1 2021.

Patients will be treated for 12 weeks, followed by a follow-up period (21 days). The total duration of participation in the study will be approximately 15 to 19 weeks from screening to the last study visit (screening and baseline could occur at the same visit). From Baseline / Day 0 onwards, randomized patients will be seen at the investigational site after 1 Week (Day 7), 2 weeks (Day 14), 4 weeks (Day 28), 8 weeks (Day 56) and 12 weeks (Day 84).

At Week 12 (Day 84 +/- 2 days), patients willing to carry on the study treatment will be able to take part in an open-label study (ABX464-302). In any other case, the subjects will exit the study (EOS) and will be treated according to the standard of care. The ABX464-302 follow-up study is a separate clinical study subject to health authorities and ethics committee approvals.

#### Study scheme:



#### 3.2 INCLUSION AND EXCLUSION CRITERIA

To be eligible for inclusion into this study, each patient must fulfil all inclusion criteria and not violate any exclusion criteria (for the protocol under which they are entered) during screening prior to randomisation.

#### 3.2.1 Inclusion criteria

A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

- Men or women age 18 75 years;
- Patient with a confirmed and documented diagnosis of adult-onset rheumatoid arthritis, for at least 12 weeks, according to the revised 2010 ACR-EULAR classification criteria, including at least one positive criteria among the following: Rheumatoid Factor (RF), Anti-Citrullinated Peptide Antibody (ACPA) or bone erosion;
- Swollen joint count of ≥ 4 (28-joint count) and tender joint count ≥4 (28-joint count) at screening;
- Patient with a moderate to severe disease activity score DAS28 CRP of ≥ 3.2 and CRP ≥ 5 mg/L (≥ 4.76 nmol)/L) at screening;



- Patient who had an inadequate response (IR), or failed either methotrexate (MTX) or/and anti-TNF $\alpha$  therapy (both administered for at least 12 weeks before IR) or were intolerant to anti-TNF $\alpha$  therapy.
  - In addition, MTX treatment should be given at a stable dose  $\geq 10$  mg/week (for at least 4 weeks prior to randomization). The maximal dose of methotrexate should not exceed a total of 20 mg/week. MTX treatment should be associated with folic acid at a dose  $\geq 5$  mg/week.

For the anti-TNF $\alpha$  therapy, the following wash-out period will be required:

- o 30 days prior to randomization for adalimumab and etanercept
- o 2 months prior to randomization for infliximab, certolizumab pegol, golimumab
- Patients with the following hematological and biochemical laboratory parameters obtained within 14 days prior to baseline:
  - Hemoglobin > 9.0 g dL-1;
  - Absolute neutrophil count ≥ 1000 mm-3;
  - Platelets  $\geq$  100,000 mm-3;
  - Total serum creatinine  $\leq 1.3 \times ULN$  (upper limit of normal);
  - Creatinine clearance > 50 mL min-1 by the Cockcroft-Gault equation within 60 days prior to baseline;
  - Total serum bilirubin < 1.5 x ULN;</li>
  - Alkaline phosphatase, AST (SGOT) and ALT (SGPT) < 1.5 x ULN;</li>
  - o Negative screening for TB and HIV, HCV, HBV
- Patients are able and willing to comply with study visits and procedures as per protocol;
- Patients should understand, sign and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures are performed;
- Patients should be affiliated to a social security regimen (for French sites only);
- Females and males receiving the study treatment and their partners must agree to use a highly effective contraceptive method during the study and for 6 months after end of study or early termination. Contraception should be in place at least 2 weeks prior to screening. Women must be surgically sterile or if of childbearing potential must use a highly effective contraceptive method. Women of childbearing potential (WOCBP) will enter the study after confirmed menstrual period and a negative pregnancy test. Highly effective methods of contraception include true abstinence, intrauterine device (IUD) or hormonal contraception aiming at inhibition of ovulation, intrauterine hormone releasing system, bilateral tubal ligation, vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the patient. In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is required. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycle. Female and male patients must not be planning pregnancy and male patients should use condom and must not donate sperm during the trial and for 6 months post completion of their participation in the trial.

## 3.2.2 Exclusion criteria

The following criteria should be checked at the time of screening. If ANY exclusion criterion applies, the patient will not be included in the study:



- Patient with a known positive anti-double stranded deoxyribonucleic acid (DNA [anti-dsDNA])
  and confirmed diagnosis of systemic lupus erythematosus (SLE);
- Patients with active infection or the following history of infection(s) (the list is not exhaustive):
  - Active infection (except benign infections, according to investigator's opinion) within 14 days prior to inclusion.
  - Serious infection, defined as an infection requiring hospitalization or IV infusion of anti-infective agents in the 2 months prior to inclusion.
  - A history of opportunistic, recurrent or chronic infections that, in the investigator's opinion, could render this study detrimental to the patient.
- Patients who have received or are expected to receive a live (including attenuated) vaccine within 3 months prior to baseline;
- Acute, chronic or history of clinically relevant (as per investigator's judgement) pulmonary, cardiovascular, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable CNS pathology such as seizure disorder, angina or cardiac arrhythmias, active malignancy or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
- Acute, chronic or history of immunodeficiency or other autoimmune disease;
- Patient previously treated with any (approved or investigational) non-anti-TNF biological disease-modifying antirheumatic drugs (bDMARDs), and targeted DMARDs (tDMARDS) prior to baseline. These treatments include: IL-6 antagonists, Janus Kinase (JAK) inhibitors, cytotoxic T lymphocyte-associated molecule CTLA-4Fc Chimera, rituximab;
- Patient treated with systemic corticosteroids >10 mg/day during the 2 weeks prior to and at randomization; IV or IM injections of glucocorticoids 4 weeks prior to randomization and IA glucocorticoids 2 weeks prior to randomization;
- Patients treated with other immunosuppressive drugs;
- History of malignancy (other than resected cutaneous basal cell or squamous cell carcinoma that
  has been treated with no evidence of recurrence) unless it has been treated and a cure is
  achieved for at least 5 years;
- Serious illness requiring systemic treatment and/or hospitalization within 3 weeks prior to baseline:
- Pregnant or breast-feeding woman;
- Illicit drug or alcohol abuse or dependency;
- Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer;
- Any condition, which in the opinion of the investigator, could compromise the patient's safety or adherence to the study protocol.



•

#### 3.3 STUDY TREATMENT

#### Medications:

- ABX464 or its matching placebo administered once daily;
- MTX ≥ 10 mg/week, at stable dose, throughout the study; the maximal dose of methotrexate should not exceed a total of 20 mg/week;
- Folic acid ≥ 5 mg/week post MTX dose, to minimize MTX toxicity.

A total of 60 patients will be recruited sequentially to receive the following doses:

| | Intervention/treatment Active Arm |
|---|---|
| Group #1 (n=20): 100mg qd | 2 capsules of 50mg ABX464 |
| Group #2 (n=20): 50mg qd | 1 capsule of 50mg ABX464 + 1 capsule of matching placebo |
| Group #3 (n=20): Placebo | 2 capsules of matching Placebo |

#### 3.4 STUDY TIMEPOINTS

Eligible patients will be enrolled in study at the screening visit within 30 days prior to the first dosing / randomization (screening and baseline could occur at the same visit, if all laboratory results are available).

Patients will be treated for 12 weeks, followed by a follow-up period (21 days).

From Baseline / Day 0 onwards, randomized patients will be seen at the investigational site after 1 Week (Day 7), 2 weeks (Day 14), 4 weeks (Day 28), 8 weeks (Day 56) and 12 weeks (Day 84).

At Week 12 (Day 84 +/- 2 days), patients willing to carry on the study treatment will be able to take part in an open-label study (ABX464-302). In any other case, the subjects will exit the study (EOS) and will be treated according to the standard of care. The ABX464-302 follow-up study is a separate clinical study subject to health authorities and ethics committee approvals.

The end of study (EOS) visit will be performed three weeks after the end of treatment period.

The total duration of participation in the study will be approximately 15 to 19 weeks from screening to the last study visit (screening and baseline could occur at the same visit).

If more than one visit occurs within a window, the nearest to the scheduled time will be presented within the summaries.

See Section 16.1 for the Study Schedule.



Visits and visit windows will be as follows:

| Visit | | Day | Window |
|-------|-----------|-----------------|----------|
| I | Screening | -30 to -1 | |
| 2 | Baseline | 0 | |
| 3 | Week I | 7 | ± 2 days |
| 4 | Week 2 | 14 | ± 2 days |
| 5 | Week 4 | 28 | ± 2 days |
| 6 | Week 8 | 56 | ± 2 days |
| 7 | Week 12 | 84 | ± 2 days |
| 8 | Week 15 | 105 (Follow-up) | ± 2 days |

## 3.5 SAMPLE SIZE CONSIDERATIONS

The primary efficacy endpoint is the rate of subjects meeting the ACR20. This response rate will be compared in subjects who received a given dose of ABX464 or placebo by likelihood ratio chi-square test. The result of the test will be interpreted in a descriptive manner therefore no adjustment for multiple comparison is applied.

For the sample size assessment, the following assumptions will be made:

- Response rate (ABX464): 0.65
- Response rate (placebo): 0.25

According to literature the ACR20 response rate for ABX464 + MTX treated subjects is expected to be between 50% and 65% while that in the placebo + MTX group is assumed to be approximately 25 to 30% (Xeljanz® Summary of Product Characteristics; ORAL Standard Investigators - N Engl J Med 2012; 367:508-519 August 9, 2012).

- Type I error: 10% two-sided
- Group allocation rate (ABX464 / placebo): I:I:I

If the above assumptions and definitions hold true with a sample size of 60 subjects receiving two doses of ABX464 or placebo in a ratio of I:I:I the study has 84% power to show a difference in response rate between one active study group and placebo.

Subjects who terminates the study prematurely will be considered failures therefore no adjustment for drop-outs is needed.

Primary safety endpoint is the rate of all treatment emergent adverse experiences. The above sample size is sufficient to detect an increase in general treatment emergent adverse experience rate from 10% to 50% with 89% power by likelihood ratio chi-square test on a 10%, two-sided significance level.



If approximately 20 subjects receive ABX464 the study has 88% chance to detect at least I specific treatment emergent AE if the underlying rate of occurrence is I:10. When the underlying rate of occurrence is around I:20 the sample size of 40 subjects receiving active treatment is sufficient to observe at least I such an event with a probability of 87% in the active treatment group.

#### 3.6 RANDOMISATION

Eligible patients (i.e. those who fulfil all inclusion/exclusion criteria) will be randomized according to a I:I:I ratio into ABX464 100mg, ABX464 50mg or placebo treatment arms.

Up to 60 patients will be randomized in this study. At the beginning, the first 6 patients will be randomized to receive either ABX464 50mg (n=4) or its matching placebo (n=2). The Data Safety Monitoring Board (DSMB) will review the safety of these first 6 patients dosed for at least 2 weeks. Once the DSMB recommendation is granted, the next patients will be randomized to receive either ABX464 50mg, ABX464 100mg or placebo. Then, a second DSMB meeting will be held after the next 6 patients are randomized to check the tolerability of the 100mg dose. Once the DSMB recommendation is granted, the next patients will be randomized to receive either ABX464 50mg, ABX464 100mg or placebo.

Randomization will be performed via a centralized treatment allocation system that will be available 24 hours-a-day, 7 days-a-week. Randomization will be stratified according to previous exposure to anti-TNF $\alpha$  therapy. The bottle numbers to be used for a specific patient will be assigned according to a predefined randomization list.

# 4 STUDY VARIABLES AND COVARIATES

## 4.1 PRIMARY VARIABLE

The primary variable for statistical comparison between treatment groups will be the incidence of treatment-emergent adverse events in the ABX464 treated Patients versus placebo, categorized by severity.

## 4.2 SECONDARY EFFICACY VARIABLES

The following secondary efficacy variables will be analysed:

## 4.2.1 Main Secondary Efficacy Endpoint

Proportion of patients achieving a categorical ACR20 response at Week 12.

The components of ACR20 assessment include:

- C-Reactive Protein (CRP) (mg/L),
- Tender/painful joint count (TJC) (28 joints),
- Swollen joint count (SJC) (28 joints),
- Patient assessment of joint pain (Pain-VAS),
- Patient global assessment of disease (PtGA),



- Physician's Global Assessment of Disease (PrGA),
- HAQ-DI

## 4.2.2 Other secondary endpoints

- Change from Baseline in the following disease parameters at Week 2, Week 4, Week 8 and Week 12:
  - Individual components of the ACR20 response (CRP, TJC(28), SJC(28), Pain-VAS, PtGA, PrGA, HAQ-DI)
  - Erythrocyte Sedimentation Rate (ESR);
  - DAS28-CRP and DAS28-ESR. The components of DAS28 assessment include TJC(28), SJC(28), CRP/ESR, and PtGA;
  - SDAI score which includes TJC(28), SJC(28), CRP, PtGA, and PrGA;
  - CDAI score which includes TJC(28), SJC(28), PtGA, and PrGA;
  - Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score
- Proportion of patients achieving at Week 2, Week 4, Week 8 and Week 12:
  - ACR20/50/70 response
  - Categorical DAS28-CRP response. Proportion of patients achieving categorical DAS28-CRP response will be measured as moderate/good European League Against Rheumatism (EULAR) response at each assessment time point;
  - Low Disease Activity (LDA) (DAS28 ≤ 3.2)
  - DAS28-ESR remission (DAS28 < 2.6)</li>
  - o ACR/EULAR remission (TJC(28), SJC(28), CRP, and PtGA: all≤1);
  - SDAI remission (SDAI  $\leq$  3.3);
  - CDAI remission (CDAI ≤ 2.8).
- Concentration of miR-124 expression in total blood (determined by qPCR) at baseline and week
- Change from Baseline in miR-124 expression in total blood at Week 8
- PK parameters:
  - o Pre-dose plasma concentration of ABX464/N-Glu at Week 2 and Week 8;
  - Post-dose plasma concentration of ABX464/N-Glu at I-, 2- and 3-hours post-dose at Baseline, Week 2 and Week 8;
  - Trough plasma concentration of ABX464/N-Glu at End of Study Visit
- The number of incidences of treatment-emergent serious adverse events;
- The number of incidences of treatment-emergent adverse events of special interest;
- The number of incidences of adverse events leading to investigational product discontinuation;
- The number of incidences of clinically significant laboratory abnormalities;
- The number of incidences of all AE (causally related and non-related) and SAE, further categorized by severity.



## 4.3 PHARMACOKINETIC VARIABLES

Pharmacokinetics will be measured via serum levels of plasma.

#### 4.4 PHARMACODYNAMIC VARIABLES

No pharmacodynamic variables will be measured.

#### 4.5 OTHER OUTCOME VARIABLES

Not applicable.

## 4.6 SAFETY VARIABLES

Safety will be evaluated by the following:

- Adverse events
- Laboratory parameters
- Vital signs (body temperature, weight, systolic and diastolic blood pressure, heart rate and respiratory rate)
- Physical examination
- ECG (PR, QRS, QT and QTc and Result: Normal, Abnormal NCS or Abnormal CS)

## 5 DEFINITIONS AND DERIVED VARIABLES

#### 5.1 DEFINITIONS

**Study Drug:** Study drug is taken to mean either ABX464 or placebo.

**Baseline:** Baseline is defined by patient and by variable as the last non-missing value before the first dose of study drug

**Study Day**: Study day is the number of days since start of treatment where the date of first dose is counted as Day 0.

**Treatment Exposure:** Treatment exposure is the number of days during the treatment period that the patient was exposed to the study treatment and is calculated as:

**Compliance:** Compliance is the number of doses actually taken divided by the scheduled number of doses expressed as a percentage.

**Non-compliance:** Non-compliance is defined as taking less than 80% or more than 120% of study medication.



**Protocol Deviation:** a deviation related to study inclusion or exclusion criteria, conduct of the trial, patient management or patient assessment. This refers to any change, divergence, or departure from the study design or procedures defined in the protocol. Deviations recorded by the Project Manager or CRA, or detected by Data Management or by Statistical programming checks as described in Section 6.3 will be identified and discussed at the Data Review Meeting before database lock to agree which should be included in Listing 16.2.2.

**Screening and enrollment:** Screening is the process of active evaluation of potential participants for enrollment in a trial. After a patient is recruited, screening occurs during the enrollment period to see if they meet the inclusion and exclusion criteria. If they meet the criteria, the subject is eligible to enroll in the trial.

**Baseline and Screening failure:** A patient is considered to be a baseline failure if the patient signs the informed consent but withdraws before the screening visit. A patient who does not fulfil the randomization criteria will be considered as a screening failure.

#### 5.2 DERIVED VARIABLES

## 5.2.1 Disease Activity Score (DAS) 28-CRP (DAS28-CRP) and DAS28-ESR

The components of the DAS28 include:

- tender/painful joint count (TJC) (28),
- swollen joint count (SJC) (28),
- CRP (in mg/L) or ESR (in mm/h), and
- patient global assessment of disease (PtGA), expressed as a Visual Analog Scale (VAS) from 0 to 100 mm

They are calculated with the following formula:

```
DAS28-CRP = 0.56 \sqrt{\text{(TJC28)}} + 0.28 \sqrt{\text{(SJC28)}} + 0.36 \text{ Ln [CRP(mg/L)} + 1] + 0.014 \text{ PtGA(VAS100mm)} + 0.96
DAS28-ESR = 0.56 \sqrt{\text{(TJC28)}} + 0.28 \sqrt{\text{(SJC28)}} + 0.70 \text{ Ln [ESR(mm/h)]} + 0.014 \text{ PtGA(VAS100mm)}
```

## 5.2.2 Simplified Disease Activity Index (SDAI)

This composite index is defined by this equation:

$$SDAI = TJC28 + SJC28 + PtGA + PrGA + CRP$$

- PtGA is expressed as a VAS from 0 to 10 cm,
- Investigator global assessment of disease (PrGA) is expressed as a VAS from 0 to 10 cm, and
- CRP (mg/L).

## 5.2.3 Clinical Disease Activity Index (CDAI)

This composite index is defined by this equation (no acute phase reactant):

$$CDAI = TJC28 + SJC28 + PtGA + PrGA$$

- PtGA is expressed as a VAS from 0 to 10 cm,
- PrGA is expressed as a VAS from 0 to 10 cm.



## 5.2.4 Categorical DAS28-CRP response

Proportion of patients achieving categorical DAS28-CRP response will be measured as moderate/good European League Against Rheumatism (EULAR) response.

The EULAR response criteria are defined as follows:

| DAS28 improvement → | > 1.2 | > 0.6 and ≤ 1.2 | ≤ 0.6 |
|---------------------|-------------------|-------------------|-------------|
| Present DAS28↓ | | | |
| ≤ 3.2 | good response | moderate response | no response |
| > 3.2 and ≤ 5.1 | moderate response | moderate response | no response |
| > 5.1 | moderate response | no response | no response |

#### 5.2.5 DAS28-ESR remission

A remission is considered when DAS28-ESR <2.6.

## 5.2.6 Low Disease Activity (LDA)

The limit to consider a Low Disease Activity (LDA) is: DAS28-ESR ≤ 3.2.

#### 5.2.7 SDAI remission

The SDAI remission is considered achieved if the SDAI score  $\leq$  3.3.

## 5.2.8 CDAI remission

The CDAI remission is considered achieved if the CDAI score  $\leq$  2.8.

## 5.2.9 ACR/EULAR remission:

In 2011, the American College of Rheumatology (ACR) and EULAR decided to set new criteria to define RA remission.

Boolean-based criteria to be used for clinical trials are:

- Tender/painful Joint Count (28)
- Swollen Joint Count (28)
- CRP
- Patient Global assessment of disease (PtGA) [VAS scale 0 10cm]

All ≤ I.

## 5.2.10 Categorical ACR20/50/70 response

The component of ACR assessment include:

- tender/painful joint count (28),
- swollen joint count (28),
- patient assessment of joint pain,
- Patient Global Assessment of Disease (PtGA)
- Physician's Global Assessment of Disease (PrGA),



- CRP and
- Disability index of the healthy assessment questionnaire (HAQ-DI).

Patient assessment of joint pain: VAS scale 0-10 cm.

**PtGA:** Patient Global Assessment of disease activity (VAS scale 0 – 10cm).

**PrGA:** Physician Global Assessment of disease activity (VAS scale 0 – 10cm).

**HAQ-DI:** This patient reported outcome questionnaire is usually self-administered by the patient.

The following 8 categories are assessed by the HAQ-DI:

- I. Dressing and grooming
- 2. Arising
- 3. Eating
- 4. Walking
- 5. Hygiene
- 6. Reach
- 7. Grip
- 8. Common daily activities

The patients report the amount of difficulty they have in performing some of these activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3).

The highest score reported by the patient for any component question of the eight categories determines the score for that category. The sum of the computed categories scores is calculated and divided by the number of categories answered. This gives a total score in the 0 to 3 range.

## **Definition of the ACR20% response:**

- ≥ 20% improvement in tender join counts
- ≥ 20% improvement swollen join counts
- ≥ 20% improvement in 3 of the 5 remaining ACR core set measures:
  - PtGA,
  - o PrGA,
  - o patient assessment of joint pain,
  - o HAQ-DI,



o CRP.

For ACR50% and ACR70%, an improvement of respectively 50 and 70% of the same parameters has to be observed.

## 5.2.11 Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue:

This questionnaire is a measure to assess the patient fatigue in chronic diseases, and is validated in RA. It includes 13 items.

The FACIT score calculation process is defined as follows:

FACIT-Fatigue Subscale Scoring Guidelines (Version 4) - Page 1

Instructions:\*

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
- 4. The higher the score, the better the QOL.

| Subscale | Item Code | Reverse it | em? | Item response | Item Sco | <u>ore</u> |
|---|---|---|---|---|---|---|
| FATIGUE | HI7 | 4 | - | | = | |
| SUBSCALE | HI12 | 4 | - | | = | |
| | An1 | 4 | - | | = | |
| | An2 | 4 | - | | = | _ |
| Score range: 0-52 | An3 | 4 | - | | = | _ |
| beore range. 0-32 | An4 | 4 | - | | = | |
| | An5 | 0 | + | | = | |
| | An7 | 0 | + | | = | |
| | An8 | 4 | - | | = | |
| | An12 | 4 | - | | = | |
| | An14 | 4 | - | | = | |
| | An15 | 4 | - | | = | |
| | An16 | 4 | - | | = | |
| | | | | Sum individual iten<br>Multipl | n scores:<br>ly by 13: | _ |
| | | | Divide | e by number of items an | swered: | =Fatigue Subscale score |

The FACIT scoring guide identifies those items that must be reversed before being added to obtain subscale totals. Negatively stated items are reversed by subtracting the response from "4". After reversing proper items, all subscale items are summed to a total, which is the subscale score. For all FACIT scales and symptom indices, the higher the score the better the QOL.

Handling missing items: If there are missing items, subscale scores can be prorated. This is done by multiplying the sum of the subscale by the number of items in the subscale, then dividing by the number of items actually answered. This can be done on the scoring guide or by using the formula below:

Prorated subscale score = Sum of item scores x N of items in subscale ÷ N of items answered

When there are missing data, prorating by subscale in this way is acceptable as long as more than 50% of the items were answered (e.g., a minimum of 4 of 7 items, 4 of 6 items, etc). The total score is then



calculated as the sum of the un-weighted subscale scores. In addition, a total score should only be calculated if ALL of the component subscales have valid scores.

## **6** ANALYSIS SETS

Membership of the analysis sets will be reviewed and agreed at a Data Review Meeting (DRM) before database lock.

#### 6.1 FULL ANALYSIS SET

The Full Analysis Set (FAS population) is defined as all patients included in the study, who have received at least one dose of the study treatment, and who have at least one baseline data.

The FAS will be used for examining demographics and other baseline characteristics. Number of doses will be presented on the FAS population.

#### 6.2 SAFETY SET

The Safety dataset (SAF population) is defined as those patients included in the study, who have received at least one dose of the study treatment.

The Safety Set will be used for all safety analyses.

#### 6.3 EFFICACY SET

## 6.3.1 "raw" Efficacy Set (Efficacy Set 1)

A "raw" efficacy set will take into consideration only patients at time point (N = nb of patients for whom efficacy variables are available at W12).

## 6.3.2 Efficacy Set with imputation (Efficacy Set 2)

Another efficacy set will use data imputation (LOCF) from Week 4.

If there are no efficacy data available, then the dropout would be considered as treatment failure.

#### 6.4 PER PROTOCOL SET

The Per Protocol dataset (PP population) is defined as those patients of the FAS population without any major protocol deviation.

Major protocol deviations are defined as deviations liable to bias the evaluation of the main efficacy endpoint. The following deviations will be considered as major (non-exhaustive list):

- Noncompliance with the inclusion or exclusion criteria;
- Noncompliance with the study treatment;



- Intake of prohibited medication;
- Noncompliance with time window.

Limited programming checks e.g. prohibited medication (based on agreed codes), lab results, may be requested and reviewed on an ongoing basis. Other potential exclusions e.g. incorrect dosing of study medication may be discussed at the DRM. The final decision on inclusion in the PP Set will be agreed and documented before database lock.

## 7 SAFETY MONITORING

An independent Data Safety Monitoring Board (DSMB), with expertise and experience in the pathology, and without direct involvement in the conduct of the trial, will be set up specifically to guarantee effective protection of patients, ensure the ethical conduct of the trial, benefit/risk ratio of the trial, and to ensure the independent review of the scientific results during the trial and at the end of the trial. Besides, the DSMB may recommend the early termination of the trial at any time if an unacceptable toxicity occurs.

The DSMB will meet after the first 6 patients are dosed (50mg or matching placebo) for at least 2 weeks to check the 50mg dose tolerability. Once the DSMB recommendation is granted, the next 6 patients will be randomized to receive either ABX464 50mg, ABX464 100mg or placebo. A second DSMB meeting will then be held when these 6 next patients are treated for at least 2 weeks, to check the 100mg dose tolerability and grant the recommendation to resume patient's randomization.

In addition, from the first DSMB onwards, meetings will be held every month during the study period. The DSMB will also review all potential causally-related Serious Adverse Events within 7 days of the initial report.

A dose limiting toxicity (DLT) is defined as a grade 3 or higher adverse event as defined by the Common Terminology Criteria for Adverse Events (CTC-AE V5.0) considered by a safety review board as probably or definitely related to study treatment. If more than 2 DLTs occur in the first 12 treated patients for at least 14 days, then the enrolment of additional patients in the treatment group will be stopped, otherwise the enrolment of planned patients will be confirmed. In addition, in case of a life threatening (grade 4) adverse reaction enrolment in the treatment group, all treatment of ongoing patients will be immediately discontinued. In both cases, enrolment will only be resumed upon the decision of the sponsor if the Data Safety Monitoring Board can conclude that the causality of the event was unrelated or unlikely related to study treatment.

The DSMB has only a consultative role. It will inform the Sponsor who will decide whether the DSMB recommendation will be followed. A DSMB charter must be available upon submission of the trial (initial protocol) to the respective competent authorities.

The sponsor will prepare the Data Safety Monitoring Board Charter which will define the primary responsibilities of the DSMB, its relationship with other study components, its members, and the purpose and timing of its meetings. The Charter will describe the process for the evaluation of dose limiting toxicities and provide the decision criteria for study continuation.



Leading up to the meeting, the data will be extracted from the EDC Database by the Database Programmer and provided to Abivax.

## 8 INTERIM ANALYSES

No interim analysis is planned.

The study analysis will be performed following database lock upon the completion of the last patient or upon its early discontinuation whichever occurs first.

## 9 DATA

#### 9.1 ECRF DATA

CRF data will be provided by Orion data management to the statistics department as SAS data sets in Orion standard format which will be used for programming the outputs to be included in the CSR. Populated data sets will be available when programming starts. These may contain dummy data if real data is not yet available.

#### 9.2 EXTERNAL DATA

## 9.2.1 Laboratory Data

Results from Local lab will be entered in CRF for Haematology, Chemistry, Pregnancy (Serum/ urine), Thyroid (for applicable sites only) and ESR (additionally for fibrinogen, troponin I & T, prothrombin time and/or INR, depending upon CSP version they get consented to).

The following table displays the clinical laboratory parameters:



| HEMATOLOGY | BIOCHEMISTRY |
|------------------------------|--------------------------------------|
| Hemoglobin | Sodium |
| Hematocrit | Potassium |
| WBC | Chloride |
| Neutrophils | Calcium |
| Lymphocytes | Phosphate |
| Monocytes | Glucose |
| Eosinophils | BUN or urea |
| Basophils | Creatinine |
| Platelet count | AST / SGOT |
| ESR | ALT / SGPT |
| Prothrombin time and/or INR* | Alkaline phosphatase |
| Fibrinogen* | GLDH |
| | LDH |
| | Lipase |
| | Total cholesterol |
| | HDL cholesterol |
| | LDL cholesterol |
| | gGT |
| | Total bilirubin |
| | Total protein |
| | Albumin |
| | CRP |
| | T3, T4, TSH ( for French sites only) |
| | Troponin I & T* |

Tests of TB (Quantiferon TB Gold Plus), HIV (anti-HIV Ab), HCV (anti-HCV Ab), HBV (HBsAg, anti-HBs Ab), anti-HCV Ab, will be performed only at screening. \* Except at Week I & 2

Reference ranges will be provided by the labs before site initiation and the required parameters will be transcribed onto the Data Management Laboratory Reference Range Form by the CRA. The CRA will provide reference ranges to the DM, who will use them to verify data on CRF. Further information or language translations will be provided by the responsible CRA if required.

A negative or positive result will be counted in the tables under number of positive or number of negative values. For a parameter with only a result in the comment stated that it is inferior to a certain value (< X), all data will be flagged where there is a sign "<" to count how many data are inferior to the detection limit.

No external data transfers are scheduled for this study.

#### 9.2.2 Other non-CRF data

There will be no other non-CRF data.

#### 9.3 RANDOMISATION LIST

The randomisation list will be uploaded to a SAS dataset following database lock.



#### 9.4 PROGRAMMING AND DATA REVIEW

Programming of analysis datasets, tables, figures and listings will be ongoing during the data management of the study. Outputs for the DSMB will be reviewed, but not fully QCd. Blind outputs may be reviewed by ABIVAX before DBL.

When the final data is considered clean, key listings (to be agreed) will be run and distributed to the study team for review. A blind data review meeting will be held to discuss the outcome of this review, the imputations for the primary endpoint and the protocol deviations. Once all data issues have been resolved and the analysis populations approved, the database will be locked. The final run of outputs and quality control (QC) will then take place.

A Data Review Meeting (DRM) may be held at the discretion of the Client. During this meeting, data listings (agreed in advance and provided by Simbec-Orion a few days before the meeting) will be used to review any outstanding problematic cases where evaluability of the data is unclear. The populations of patients for the statistical analysis and reporting of the study will be agreed and recorded by the study Statistician.

The study Data Manager, Statistician or Statistical Programmer, Project Manager and a Medic of Simbec-Orion will attend the DRM with representatives of Abivax.

## 10 STATISTICAL METHODS

#### 10.1 GENERAL PRINCIPLES

All statistical methods will be based on the International Conference on Harmonisation (ICH) E9 document "Statistical Principles for Clinical Trials".

Data will be summarised by treatment group. A total column showing all patients will be included for baseline and safety summaries. Where appropriate, data will also be summarised by visit with summaries for each visit attended as scheduled and an additional summary for final (last scheduled visit or early withdrawal). The format of the summaries is defined in the shells at the end of this document.

In summary and analysis tables of continuous variables, standard descriptive statistics (N, mean, standard deviation [SD], median, minimum and maximum) will be presented. Least squares mean (LS mean), standard error (SE) and 95% confidence interval (CI) will be presented in the statistical analysis outputs as appropriate. For PK summaries, arithmetic mean (AM), geometric mean (GM) and coefficient of variation (%CV) will be used to summarise the data. The minimum and maximum statistics will be presented in summary tables to the same number of significant figures as the original data. The mean/AM, median, LS mean, GM, CI, SD and SE will be presented to one more significant than the original data.

For numeric data which includes non-numeric values (e.g. PK data reported as Below Limit of Qualification (BLQ) or lab results reported as < 10 or >100) the following principles will be applied when summarising the data:



- BLQ will be replaced with a value that is ½ of the lower limit of quantification (LLQ);
- Results reported as < x will be treated in the same way as BLQ with LLQ=x;</li>
- Otherwise AM, GM, SD, Cl and %CV will not be calculated;
- Whenever meaningful, minimum, median and maximum will be presented based on the reported data (e.g. minimum = <10, median = 20, maximum = >100).

In summary tables of categorical variables, the number of non-missing observations by category will be presented with percentages. The number of missing observations will also be presented when non-zero. Unless otherwise specified, the denominator for each percentage will be the number of non-missing observations within the column. All percentages will be presented to one decimal place.

Patient line plots will use actual time on the time axis. Mean plots will use a linear time scale for the nominal times of the visits and will be labelled by visit. Results from an early withdrawal visit will be excluded.

If changes in severity for the same TEAE have been reported separately but with the same AE number, they will be collapsed to a single AE with maximum severity for the summary tables, but listed as reported.

Classifications of medical history, concomitant medication and adverse events will be sorted alphabetically within the summary tables.

If any laboratory assessments are repeated at the same visit, the result from the repeat assessment will be used in summaries. Both values will be listed.

CRF data collected/ Data collected on the eCRF will be presented within data listings. The data listings will be sorted by treatment group, country, centre number, patient number and visit/week/day. Treatment group will be as allocated (randomised). If any patients receive the wrong treatment this will be flagged in all listings. Visits outside the visit windows will be identified within the listings. For patients who complete the study, the last visit will be described in the listings as '<Day X>'; for those who withdraw early it will be described as 'End of Study'.

The date format for all output presentations will be 'ddMMMyyyy'.

All statistical analysis will be performed using SAS 9.2 or higher.

All hypothesis testing will be carried out at the 5% (2-sided) significance level unless stated otherwise.

P-values will be rounded to four decimal places. P-values less than 0.0001 will be reported as <0.0001 in tables.

If any of the assumptions underlying the formal statistical methods proposed are violated during the analysis of the final data, alternative statistical methods will be used and any changes documented in the statistical methods section of the clinical study report (CSR), including the rationale for use.



#### 10.2 STRATIFICATION AND COVARIATE ADJUSTMENT

Randomization will be stratified according to a single factor: patients without previous exposure to anti-TNF $\alpha$  therapy versus patients with previous exposure to anti-TNF $\alpha$ .

#### **10.3** Interactions

The interaction between treatment in two different doses and placebo will be investigated for the primary endpoint (incidence of treatment-emergent adverse events categorized by severity).

#### 10.4 MISSING DATA

For total scores and subscales with missing items the following rule will be used:

If < 50% of the scale items are missing, the total (or subscale total) will be calculated using the mean score of the non-missing items for that scale or subscale to impute a score for the missing items. In practice the score is derived using the formula:

total of non-missing items x number of items in (sub)scale / number of non-missing items

If > 50% of the items were missing, no scale or subscale score will be calculated; the score will be considered missing.

There will be no other imputation of missing data in this study.

## 10.5 POOLING OF SITES

Sites will be pooled for all analyses. There will be no adjustment for centre effect or treatment by centre interaction.

#### 10.6 MULTIPLE COMPARISONS

There will be no corrections to nominal p-values for multiple comparisons because the results of the tests will be interpreted in a descriptive manner.

## 10.7 SUBGROUP ANALYSES

Not applicable.

#### 10.8 STATISTICAL ISSUES

Not applicable.



## 11 STATISTICAL OUTPUT

General principles for layout of the statistical output are described in Section 10.1, including specification of the table columns, and these are illustrated for each unique table in the table shells in Section 15. For clarity and brevity in this document the phrase "by treatment group" is understood for all summaries and is not included within the text of this section.

#### 11.1 PATIENT DISPOSITION

A summary of the number of screened patients, baseline failures, screening failures and reasons for screening failure will be produced for all enrolled patients (*Table 14.1.1*). The patient disposition table (*Table 14.1.2*) will summarise the following data for all randomised patients:

- The number (%) of patients in the FAS,
- The number (%) of patients in the Safety Set,
- The number (%) of patients in the PP Set.

The number (%) of patients who withdraw from the study and the main reason for withdrawal will be summarised. (*Table 14.1.3*)

A listing of all patients with protocol deviations will be presented. A data listing presenting the eligibility for the analysis sets for each patient will also be presented.

#### 11.2 PATIENT CHARACTERISTICS AT BASELINE

## 11.2.1 Demographic and Baseline Characteristics

Demographics and other baseline characteristics will be summarized by treatment arm (*Table 14.1.4*). This analysis will be conducted on the FAS population.

Age will be calculated using Date of Birth (DOB) and Date of first treatment (Visit I) and presented as age at last birthday as an integer.

BMI is the patient's body weight in kilograms divided by the square of the patient's height in metres.

## 11.2.2 Medical History and Current Medical Conditions

All conditions will be coded using the version 23.0 of the Medical Dictionary for regulatory Activities (MedDRA) defined in the Data Management Plan. Past medical/surgical history and current medical conditions will be summarised by system organ class (SOC) and preferred term (PT). The number (%) of patients reporting each condition will be presented using the FAS (*Table 14.1.5.1 and 14.1.5.2*).

#### 11.3 EFFICACY ANALYSES

Analysis of efficacy data will be carried out on Efficacy Set I and will be repeated for Efficacy Set 2. Treatment comparisons will be ABX464 in two different doses vs. placebo.



## 11.3.1 Primary Variable

The primary efficacy endpoint of the study, the ACR20 response rate, will be compared in subjects who received a given dose of ABX464 or placebo by likelihood ratio chi-square test on a 10% two-sided level (Table 14.2.1.1 and Table 14.2.1.2).

The result of the test will be interpreted in a descriptive manner therefore no adjustment for multiple comparison is applied.

## 11.3.2 Secondary Variables

Descriptive statistics will be presented by treatment arm for all secondary efficacy variables for each measurement timepoints separately for the study groups:

- Proportion of patients achieving a categorical ACR20 response at Week 12 (*Table 14.2.2.1* and *Table 14.2.2.2*).
- Change from Baseline in the individual components of the ACR20 response at Week 2, Week 4, Week 8 and Week 12 (*Table 14.2.3.1* and *Table 14.2.3.2*):
  - o C-Reactive Protein (CRP) (mg/L),
  - o Tender/painful joint count (TJC) (28 joints),
  - Swollen joint count (SJC) (28 joints),
  - Patient assessment of joint pain (Pain-VAS),
  - o Patient global assessment of disease (PtGA),
  - Physician's Global Assessment of Disease (PrGA),
  - o HAQ-DI.
- Change from Baseline in the following disease parameters at Week 2, Week 4, Week 8 and Week 12:
  - o ESR (Table 14.2.4.1.1 and Table 14.2.4.1.2);
  - DAS28-CRP (Table 14.2.4.2.1 and Table 14.2.4.2.2) and DAS28-ESR (Table 14.2.4.3.1 and Table 14.2.4.3.2);
  - SDAI score (Table 14.2.4.4.1 and Table 14.2.4.4.2);
  - CDAI score (Table 14.2.4.5.1 and Table 14.2.4.5.2);
  - o FACIT-Fatigue score (Table 14.2.4.6.1 and Table 14.2.4.6.2).
- Proportion of patients achieving:
  - ACR20/50/70 response;
  - Categorical DAS28-CRP response;
  - o LDA;
  - DAS28-ESR remission;
  - ACR/EULAR remission;
  - SDAI remission;
  - CDAI remission

at Week 2, Week 4, Week 8 and Week 12 (Table 14.2.5.1 and Table 14.2.5.2).

These statistics include:



- Continuous variables: mean, standard deviation, minimum and maximum, stratified 95% confidence intervals, median and quartiles will be presented.
- Categorical variables: counts, rates and stratified 95% confidence intervals for the rates will be calculated.

In addition to descriptive statistics, mixed model analysis of covariance will be conducted for the following measurements:

- The change from baseline in DAS28-CRP and DAS28-ESR;
- The change from baseline in the individual components of the ACR20 response (CRP, TJC(28), SJC(28), Pain-VAS, PtGA, PrGA, HAQ-DI) and in ESR;
- The change from baseline in SDAI and CDAI scores.

In this model, treatments and stratum will be fixed effects, subjects will be random effect, and baseline values of the respective measurements will be covariates. Other explanatory variables will also be allowed to be included in the model. In order to normalize eventual skewed distributions transformation of the data will also be considered. Study groups will be compared within this model framework. All p-values will be interpreted in a descriptive manner.

All other analyses will be descriptive.

## 11.4 PK ANALYSES

PK analysis will not be conducted by Simbec-Orion.

## 11.5 PD ANALYSES

Not applicable.

#### 11.6 SAFETY ANALYSES

## 11.6.1 Adverse Events

An overall summary table will be presented (any adverse event, any treatment emergent adverse event (TEAE), any serious adverse event (SAE), death, any grade 3 or higher adverse events from baseline to the end of Study) (*Table 14.3.1.1*). This analysis will be conducted on SAF population.

Primary safety endpoint, the rate of all treatment emergent adverse experiences, will be compared in subjects who received a given dose of ABX464 or placebo by likelihood ratio chi-square test on a 10% two-sided significance level (14.3.1.2.1).

Two periods will be defined for TEAE:

- Period I: any adverse event which occurs or worsens from first dosing to Day 84;
- Period II: any adverse event which occurs after Day 84.



Adverse events will be described by primary system organ class and preferred term according to the two periods. Numbers and percentage of patients, and number of occurrences of adverse event will be presented for:

- TEAE (Table 14.3.1.2.2 and Table Table 14.3.1.2.3);
- Serious TEAE (Table 14.3.1.3.1 and Table Table 14.3.1.3.2);
- TEAE leading to drug discontinuation (*Table 14.3.1.4.1* and *Table Table 14.3.1.4.2*);
- TEAE of grade 3 or 4 (Table 14.3.1.5.1 and Table Table 14.3.1.5.2);

Further assessment of safety will be based on the frequency of adverse events (with and without regard to causality) graded according to the CTC-AE Classification and also, the review of individual values for clinical laboratory data, vital signs and ECG focusing on the detection of abnormal values and PCSAs [potentially clinically significant abnormalities (PCSAs) determined upon investigator considerations].

Adverse events will be tabulated (counts and percentages) by group. All adverse events will be listed, and the data will be tabulated by body system/organ class. Adverse event tabulations will include all treatment emergent adverse events, which will be further classified by severity, and relationship to treatment and dose level.

All adverse events (AE) will be classified using the version of the MedDRA coding dictionary specified in the DHM.

Events will be classified as treatment-emergent if they started or increased in severity on or after the first date and time of medication dosing at Visit I and up to study closure or withdrawal date. If an event start date is partial, then the start day, month, year or stop date will be used to determine if the event is treatment-emergent. If the classification of the AE cannot be determined from the data available, then the event will be considered treatment-emergent.

Treatment-emergent adverse events (TEAEs) will be further classified as follows:

Severe TEAEs: Severity classified as 'severe' (Common Toxicity Criteria [CTC] grade 3 or 4) or missing.

Serious TEAEs: Serious classified as 'yes' or missing.

Drug-related TEAEs: Relationship to study drug classified as 'related' or missing.

**Serious drug-related TEAEs**: Both serious and drug-related, as specified above.

TEAEs leading to withdrawal from study: Action taken classified as 'discontinued'.

All AE summary tables will show the number (%) of patients having at least one event and the number of events in each treatment group and overall. Median duration of AEs (from baseline to occurrence) will be presented in the tables. Note: If a patient has multiple AEs with the same preferred term, these will be summarised once within the count for N (%) of patients, but each event will be counted within the number of reports n of each AE. Changes in severity of the same AE (if collected) will be counted only once within the number of reports n of each AE.

The following will be presented in listing format within the data summaries:

• Deaths (*Table 14.3.2.1*);



- Serious Adverse Events (Table 14.3.2.2);
- Adverse Events which Led to Withdrawal (*Table 14.3.2.3*).

All adverse events (including non-treatment-emergent events) recorded on the CRF will be listed within the data listings.

## 11.6.2 Laboratory Data

For hematology and biochemistry panels, local laboratory will be used.

Descriptive statistics (n, mean, SD, SEM, median, minimum and maximum) for laboratory parameters will be computed at each scheduled assessment (*Table 14.3.3.1 and Table 14.3.3.2*). If relevant for some parameter, change from baseline will also be tabulated.

Each laboratory value that is outside of the institution's normal range will be identified. The Investigator will be responsible for assessing the clinical significance of laboratory abnormalities. If the Investigator is uncertain about the clinical significance of a laboratory abnormality, he/she will consult with the Sponsor medical monitor.

Laboratory data listings will be presented in two ways:

- Abnormal values (presented within the data summaries) (Table 14.3.3.3)
- All laboratory data (presented within the data listings)

The absolute values of each parameter will be summarised at each visit.

In addition, shift tables from baseline will be presented.

If lab results are repeated at the same visit, the repeated result will be used in summaries (instead of the original one) provided the sample was taken within the visit window, otherwise the original result will be used. All results will be listed.

Lab results at unscheduled visits will be included in the listings but will not be summarised.

Serum pregnancy data will be listed only.

## 11.6.3 Vital Signs

Vital signs will be summarized by using descriptive statistics (n, mean, SD, SEM, median, minimum and maximum) (*Table 14.3.4*). Number of patients with at least one abnormal value will be tabulated (counts and percentages) for each parameter in summary shift tables, by group and dose.

Measurements of vital signs will be done at each visit (Blood pressure, Heart Rate, Body temperature).

The investigator should ensure that each parameter outside the normal range is assessed for clinical significance. For any deviation assessed clinically significant, the investigator has to document the change as an AE in the CRF.

In addition, it is at the discretion of the investigator to document any change or trend over time in vital signs as an AE if he considers the change to be clinically significant, even if the absolute value is within the alert limit or reference range.



## 11.6.4 Physical Examination

A routine physical examination (including body weight) will be done at each study visit. Physical examinations will cover eyes, ears, nose, throat, lungs/thorax, heart/cardiovascular system, abdomen, skin and mucosae, nervous system, lymph nodes, musculo-skeletal system, and, if applicable, others. Any new clinically relevant finding compared to baseline must be documented as adverse event.

Shift tables will be presented showing changes from baseline to each visit for normal / abnormal physical examination results (*Table 14.3.5*).

## 11.6.5 Electrocardiogram

Electrocardiograms will be performed at Screening, Baseline / Day 0, Week 8 / Day 56 and at the EOS visit (in case of premature discontinuation only). At least a 12-lead ECG with recordings of at least 6 action potentials in lead II (paper speed 25mm/s, amplitude 10mm/mV) will be measured at a resting position. Resting ECG should be performed before any examinations.

All abnormal findings must be documented in the CRF. Any clinically relevant findings compared to ECG done at Day 0 / Baseline must be documented as adverse events.

The absolute values of PR, QRS, QT and QTc will be summarised at each visit done (screening, baseline, week 8 and EOS) (*Table 14.3.6*).

The number and percentage of the patients with Normal / Abnormal NCS / Abnormal CS ECG results will be summarised.

## 11.7 STUDY DRUG EXPOSURE AND COMPLIANCE

Treatment exposure (ABX464 50mg, 100mg or placebo) and compliance (yes/no) will be summarised for the FAS (*Table 14.3.7*).

## 11.8 PRIOR AND CONCOMITANT MEDICATION

All medications taken by patients on entry to the study or during the study will be recorded in the CRF. Medications will be classified using the version of the World Health Organisation Drug Dictionary (WHODD) coding dictionary defined in the Data Management Plan. The Anatomical Therapeutic Chemical (ATC) Classification and WHO-DRUG PT will be used to list and summarise the data.

If required by client, conmeds can be summarised at 3 levels: ATC levels 1 and 2 and preferred term.

**Prior medications** are defined as medication that started and stopped before Day I. Only medications where the stop date is prior to Day I will be considered prior. If the stop date is unknown or incomplete and the medications cannot definitely be considered as stopped prior to Day I then the medications will be considered as concomitant medications at randomisation or change in concomitant medication, depending on the start date.

**Concomitant medications at randomisation** are defined as medications that started before Day I and either stopped on Day I or continued into the study. Partial start dates where the medication cannot



definitely be considered as starting prior to Day I will lead to a categorisation of the medications as having started on or after dosing.

**Change in concomitant medication** is defined as medication that started on or after Day I. If the medication start or stop dates are partial then the rules for prior and concomitant medication, detailed above will be observed prior to assigning a category.

The number (%) of patients reporting the use of any prior medications and the number (%) of patients taking each drug by ATC classification and PT will be summarised using the FAS (*Table 14.3.8*). This table will be repeated for concomitant medications at randomisation (*Table 14.3.9.1*) and for change in concomitant medication (*Table 14.3.9.2*)

## Mandatory concomitant treatments are the followings:

- MTX ≥ 10 mg/week, at stable dose, throughout the study;
- Folic acid ≥ 10 mg/week post MTX dose, to minimize MTX toxicity.

## **Allowed Concomitant Medications are the followings:**

- Corticosteroids at stable dose of prednisone and prednisone equivalent ≤10 mg/day during the study;
- Non-steroidal anti-inflammatory drugs (NSAIDs) at stable dose during the study;
- Antalgics including class III at stable dose during the study;
- Other non-rheumatologic medications.

Potential other concomitant medications (not indicated for rheumatoid arthritis) should be kept at constant dose during the course of the study and properly reported in the medical file of the patient and the eCRF.

## Prohibited concurrent medications are the followings:

- Any non-anti-TNFα biological or targeted DMARDs: IL-6 antagonists, JAK inhibitors, CTLA-4Fc Chimera, rituximab;
- Any immunosuppressive drugs;
- Vaccination with live components during the study and up to 8 Weeks after the last dosing;
- Drugs that could interact with ABX464 should be avoided especially the CYPIA2 substrates.
  The following CYPIA2 substrates with a narrow therapeutic margin are prohibited during the
  whole course of the study (rifampicin, clozapine, theophylline, ropinirole, warfarin and
  methadone). In case of concomitant treatment with ondansetron, the maximal daily dose must
  be limited to 8 mg;
- Use of any investigational or non-registered product within 3 months preceding baseline.



## 12 VALIDATION

All tables, figures and listings will be subject to independent quality control and visual review. Unique tables will be independently programmed. Findings will be documented in a quality control form and actions taken will also be documented.

The completed form will be reviewed and signed by both programmers and by the head of biostatistics.

# 13 LITERATURE CITATIONS/REFERENCES

Not applicable


## 14 LIST OF TABLES, FIGURES AND LISTINGS

#### 14.1 LIST OF TABLES

## Demographic Data

| Table 14.1.1 | Screening Failures | All Enrolled Patients |
|---|---|---|
| Table 14.1.2 | Patient Disposition | All Randomised Patients |
| Table 14.1.3 | Study Termination and Primary Reason for Withdrawal | All Randomised Patients |
| Table 14.1.4 | Demographic and Baseline Characteristics | Full Analysis Set |
| Table 14.1.5.1 | Medical History | Full Analysis Set |
| Table 14.1.5.2 | Current Medical Conditions | Full Analysis Set |

#### Efficacy Data

| Efficacy Set 1 |
|----------------|
| Efficacy Set 2 |
| PP Set |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |
| Efficacy Set 2 |
| Efficacy Set 1 |



| Table 14.2.4.5.2 | Analysis of CDAI Score | Efficacy Set 2 |
|---|---|---|
| Table 14.2.4.6.1 | Summary of FACIT-Fatigue Score | Efficacy Set 1 |
| Table 14.2.4.6.2 | Summary of FACIT-Fatigue Score | Efficacy Set 2 |
| Table 14.2.5.1 | Summary of Patients Different Responses and Remissions | Efficacy Set 1 |
| Table 14.2.5.2 | Summary of Patients Different Responses and Remissions | Efficacy Set 2 |

## Safety Data

| Table 14.3.1.1 | Summary of Adverse Events | Safety Set |
|---|---|---|
| Table 14.3.1.2.1 | Analysis of all Treatment-Emergent Adverse Events | Safety Set |
| Table 14.3.1.2.2 | Treatment-Emergent Adverse Events, by SOC and PT: Period I | Safety Set |
| Table 14.3.1.2.3 | Treatment-Emergent Adverse Events, by SOC and PT: Period 2 | Safety Set |
| Table 14.3.1.3.1 | Serious Treatment-Emergent Adverse Events, by SOC and PT: Period 1 | Safety Set |
| Table 14.3.1.3.2 | Serious Treatment-Emergent Adverse Events, by SOC and PT: Period 2 | Safety Set |
| Table 14.3.1.4.1 | Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation, by SOC and PT: Period I | Safety Set |
| Table 14.3.1.4.2 | Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation, by SOC and PT: Period 2 | Safety Set |
| Table 14.3.1.5.1 | Treatment-Emergent Adverse Events of Grade 3 or 4 by SOC and PT: Period I | Safety Set |
| Table 14.3.1.5.2 | Treatment-Emergent Adverse Events of Grade 3 or 4 by SOC and PT: Period 2 | Safety Set |
| Table 14.3.2.1 | Listing of Deaths | Safety Set |
| Table 14.3.2.2 | Listing of Serious Adverse Events | Safety Set |
| Table 14.3.2.3 | Listing of Withdrawals Due to Adverse Events | Safety Set |
| Table 14.3.3.1 | Summary of Laboratory Parameters: Haematology | Safety Set |
| Table 14.3.3.2 | Summary of Laboratory Parameters: Biochemistry | Safety Set |
| Table 14.3.3.3 | Listing of Abnormal Laboratory Values | Safety Set |
| Table 14.3.4 | Vital Signs | Safety Set |
| Table 14.3.5 | Shift Table of Physical Examination | Safety Set |
| Table 14.3.6 | Electrocardiogram | Safety Set |
| Table 14.3.7 | Study Drug Exposure and Compliance | Full Analysis Set |



| Table 14.3.8 | Prior Medications | Full Analysis Set |
|----------------|------------------------------------|-------------------|
| Table 14.3.9.1 | Concomitant Medications | Full Analysis Set |
| Table 14.3.9.2 | Changes in Concomitant Medications | Full Analysis Set |

#### 14.2 LIST OF LISTINGS

## Patient Data Listings

| Listing 16.2.1.1 | Patient Disposition |
|------------------|----------------------------------------------|
| Listing 16.2.1.2 | Discontinued Patients |
| Listing 16.2.2 | Protocol Deviations |
| Listing 16.2.3 | Analysis Datasets |
| Listing 16.2.4 | Demographic Data |
| Listing 16.2.5 | Study Drug Exposure and Compliance |
| Listing 16.2.6 | Efficacy Response Data: ACR20/50/70 Response |
| Listing 16.2.7 | Adverse Event Listing |
| Listing 16.2.8.1 | Laboratory Measurements: Haematology |
| Listing 16.2.8.2 | Laboratory Measurements: Biochemistry |

# Individual Patient Data Listings (Archive)

| Listing 16.4.1 | Final Status |
|---|---|
| Listing 16.4.2 | Patient Visit Dates |
| Listing 16.4.3.1 | Inclusion Criteria |
| Listing 16.4.3.2 | Exclusion Criteria |
| Listing 16.4.4 | Medical History |
| Listing 16.4.5.1 | Raw Efficacy Data: Individual Components of the ACR20 Response |
| Listing 16.4.5.2 | Raw Efficacy Data: ESR, DAS28-CRP, DAS28-ESR, SDAI Score, CDAI Score and FACIT-Fatigue Score |
| Listing 16.4.5.3 | Raw Efficacy Data: Different Responses and Remissions |
| Listing 16.4.9 | Vital Signs |
| Listing 16.4.10 | Physical Examination |
| Listing 16.4.11 | 12-Lead Electrocardiogram |
| Listing 16.4.12.1 | Prior Medications |



| Listing 16.4.12.2 | Concomitant Medications |
|-------------------|-------------------------------|
| Listing 16.4.12.3 | Changes to Medications |
| Listing 16.4.13 | Pregnancy Test |
| Listing 16.4.14 | Laboratory Samples Collection |

## 15 SHELLS FOR TABLES, FIGURES AND LISTINGS

The intended layouts for tables, figures and listings are presented. However, it may be appropriate for the Orion programmer to change the layouts, upon review of the data available, for completeness and clarity.

QCd output will be produced as Rich Text Format (.rtf) files for convenient inclusion in the CSR.

Subject to this, the following will apply:

- Layout will be landscape, fixed width, font size 8.
- Each output will have the heading:
   ABX464-301 (left); date ddMMMyyyy (right)
- Table headings will define the analysis set used for the summary/analysis.
- All outputs will have a footer specifying the SAS program path and filename (left); page x/y (right)
- Tables will have a footer specifying the source listing
- · Figures will have a footer specifying the source table or listing
- Additional footnotes will be included where appropriate for clarification.
- Treatment group and patient number and will be included in all listings.



| | Total Enrolled | |
|---|---|---|
| | (N=xx) | |
| Total number of enrolled patients | xx | |
| Screened | xx (xx.x%) | |
| Randomised | xx (xx.x%) | |
| Screening failure | xx (xx.x%) | |
| Baseline failure | Xx (xx.x%) | |
| Primary Reason for screening failure | | |
| Inclusion criterion not met | xx (xx.x%) | |
| Exclusion criterion | xx (xx.x%) | |
| Withdrawal by patient | xx (xx.x%) | |
| Etc | | |
| he denominator for each percentage is the number of enroll | ed patients. | |
| ource: Listing 16.2.1.1 and 16.2.1.2 | | |
| ath\Filename | | Page x/y |



| | Table 14.1.2 Patio | ent Disposition (All Rar | l Randomised Patients) | |
|---|---|---|---|---|
| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
| Full Analysis Set | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Safety Set | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Efficacy Set 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Efficacy Set 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Per Protocol Set | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

The denominator for each percentage is the number of randomized patients in the column.

Source: Listing 16.2.1.1 and 16.2.1.2

Path\Filename



Table 14.1.3 Study Termination and Primary Reason for Withdrawal (All Randomised Patients)

| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Randomised | xx | xx | xx | xx |
| Completed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Early withdrawal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Main reason for early withdrawal | | | | |
| Investigator's decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Major protocol violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patient's decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal of consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

The denominator for each percentage is the number of randomized patients in the column. Completed defined as performed follow-up visit.

Source: Listing 16.2.1.1 and 16.2.1.2

Path\Filename



ABX464-301

ddMMMyyyy
Table 14.1.4 Demographic and Baseline Characteristics (Full Analysis Set)

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464 | Placebo | Total |
|---|---|---|---|---|---|
| | | | 50mg | (N=xx) | (N=xx) |
| | | | (N=xx) | (N-XX) | (14-88) |
| age (years) | N | XX | xx | xx | xx |
| , | Mean | xx.xx | xx.xx | xx.xx | XX.XX |
| | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | xx.xx | xx.xx | xx.xx | XX.XX |
| | Minimum | xx.x | xx.x | xx.x | XX.X |
| | Maximum | xx.x | xx.x | xx.x | xx.x |
| sex | N | xx | xx | xx | xx |
| | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Height (cm) | N | xx | xx | xx | xx |
| | Mean | xx.xx | xx.xx | xx.xx | XX.XX |
| | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | xx.xx | xx.xx | xx.xx | XX.XX |
| | Minimum | xx.x | xx.x | xx.x | XX.X |
| | Maximum | xx.x | xx.x | xx.x | xx.x |
| Weight (kg) | N | xx | xx | xx | xx |
| | Mean | xx.xx | xx.xx | xx.xx | XX.XX |
| | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | xx.xx | xx.xx | xx.xx | XX.XX |
| | Minimum | xx.x | xx.x | xx.x | XX.X |
| | Maximum | XX.X | xx.x | xx.x | xx.x |
| BMI (kg/m2) | N | xx | xx | xx | xx |
| | Mean | xx.xx | xx.xx | xx.xx | XX.XX |



| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| SD | xx.xx | xx.xx | xx.xx | xx.xx |
| Median<br>Minimum | xx.xx<br>xx.x | xx.xx<br>xx.x | xx.xx<br>xx.x | xx.xx<br>xx.x |
| Maximum | xx.x | XX.X | XX.X | xx.x |

The denominator for each percentage is the number of non-missing observations within the column Age was calculated using DOB and date of first treatment (Visit 1) and presented as age at last birthday. BMI is the patient's body weight in kilograms divided by the square of the patient's height in metres.

Source: Listing 16.2.4

Path\Filename



ABX464-301

Table 14.1.5.1 Medical History (Full Analysis Set)

ddMMMyyyy

| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| any medical/surgical history | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 50C | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 50C | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Etc

The denominator for each percentage is the number of patients within the column.

Medical history refers to conditions which stopped prior to or at the screening visit.

Source: Listing 16.4.4

Path\Filename

Page x/y

This layout also applies to:

Table 14.1.5.2 Current Medical Conditions (Full Analysis Set) [Programmer's Note: Update footnote to medical conditions definition.]



Table 14.2.1.1 Analysis of ACR20 Response Rate (Efficacy Set 1)

| | | ABX-464<br>100mg<br>(N=xx) | 100mg 50mg | | p-value |
|---|---|---|---|---|---|
| ACR20 Response | N | xx | xx | xx | |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Response rate between treatments is compared using likelihood ratio chi-square test at a two-sided 10% significance level.

Source: Listing 16.2.6

Path\Filename

Page x/y

This layout also applies to:
Table 14.2.1.2 Analysis of ACR20 Response Rate (Efficacy Set 2)
Table 14.2.1.3 Analysis of ACR20 Response Rate (PP Set)



Table 14.2.2.1 Summary of Categorical ACR20 Response at Week 12 (Efficacy Set 1)

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Week 12 | N | xx | xx | xx |
| | Rate | xx.x % | xx.x % | xx.x % |
| | Stratified 95% CI | xx.x % - xx.x % | xx.x % - xx.x % | xx.x % - xx.x % |

Source: Listing 16.2.6

Path\Filename

Page x/y

This layout also applies to:

Table 14.2.2.2 Summary of Categorical ACR20 Response at Week 12 (Efficacy Set 2)



Table 14.2.3.1 Analysis of the individual components of the ACR20 response (Efficacy Set 1)

| | | ABX-464 | ABX-464 | Placebo | |
|---|---|---|---|---|---|
| | | 100mg | 50mg | (N=xx) | p-value |
| | | (N=xx) | (N=xx) | (N-XX) | |
| P | | | | | |
| Baseline | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean | xx.xx | XX.XX | XX.XX | |
| | Stratified 95% CI | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx | |
| | SD | xx.xx | XX.XX | XX.XX | |
| | Minimum | xx.x | XX.X | XX.X | |
| | Maximum | xx.x | XX.X | XX.X | |
| | Median | xx.xx | XX.XX | XX.XX | |
| | Quartiles | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx | |
| Week 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean | xx.xx | xx.xx | xx.xx | |
| | Etc | | | | |
| Change from baseline to Week 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| emange tram susceed to meek = | Mean | XX.XX | XX.XX | XX.XX | |
| | Etc | ,,,,,, | | AAAAA | |
| Analysis of Covariance (change from baseline to Week 2) | | | | | x.xxxx |
| Week 4 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean<br>Etc | xx.xx | xx.xx | xx.xx | |
| Etc | | | | | |



Etc

Mixed model analysis of covariance is conducted for the changes of baseline for each parameter.

Source: Listing 16.4.5.1

Path\Filename

Page x/y

Programmer's Note: list of variables consists of CRP, TJC, SJC, Pain-VAS, PtGA, PrGA, HAQ-DI.

This layout also applies to:

Table 14.2.3.2 Analysis of the individual components of the ACR20 response (Efficacy Set 2)



ABX464-301

#### Table 14.2.4.1.1 Analysis of ESR (Efficacy Set 1)

ddMMMyyyy

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | p-value |
|---|---|---|---|---|---|
| Baseline | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean | xx.xx | XX.XX | XX.XX | |
| | Stratified 95% CI | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx | |
| | SD | xx.xx | XX.XX | XX.XX | |
| | Minimum | xx.x | XX.X | XX.X | |
| | Maximum | xx.x | XX.X | XX.X | |
| | Median | xx.xx | XX.XX | XX.XX | |
| | Quartiles | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx | |
| week 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean | xx.xx | XX.XX | XX.XX | |
| | Etc | | | | |
| Change from baseline to Week 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean | xx.xx | xx.xx | xx.xx | |
| | Etc | | | | |
| Analysis of Covariance (change from baseline to Week 2) | | | | | x.xxxx |
| to also d | N | / 9/ | / 9/\ | / 9/ | |
| Week 4 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | |
| | Mean<br>Etc | xx.xx | XX.XX | XX.XX | |
| Etc | | | | | |



Mixed model analysis of covariance is conducted for the changes of baseline for each parameter.

Source: Listing 16.4.5.2

Path\Filename

```
This layout also applies to:

Table 14.2.4.1.2 Analysis of ESR (Efficacy Set 2)

Table 14.2.4.2.1 Analysis of DAS28-CRP (Efficacy Set 1)

Table 14.2.4.2.2 Analysis of DAS28-CRP (Efficacy Set 2)

Table 14.2.4.3.1 Analysis of DAS28-ESR (Efficacy Set 1)

Table 14.2.4.3.2 Analysis of DAS28-ESR (Efficacy Set 2)

Table 14.2.4.4.1 Analysis of SDAI Score (Efficacy Set 1)

Table 14.2.4.4.2 Analysis of SDAI Score (Efficacy Set 2)

Table 14.2.4.5.1 Analysis of CDAI Score (Efficacy Set 1)

Table 14.2.4.5.2 Analysis of CDAI Score (Efficacy Set 2)
```



| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Baseline | N | | | vv (vv v %) |
| Baseline | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Mean | xx.xx | xx.xx | XX.XX |
| | Stratified 95% CI | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx |
| | SD | xx.xx | XX.XX | xx.xx |
| | Minimum | xx.x | xx.x | xx.x |
| | Maximum | xx.x | xx.x | xx.x |
| | Median | xx.xx | xx.xx | xx.xx |
| | Quartiles | xx.xx - xx.xx | xx.xx - xx.xx | xx.xx - xx.xx |
| Neek 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Mean | xx.xx | xx.xx | xx.xx |
| | Etc | | | |
| Change from baseline to Week 2 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| - | Mean | xx.xx | xx.xx | xx.xx |
| | Etc | | | |
| Neek 4 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Mean | xx.xx | xx.xx | XX.XX |
| | Etc | | | |
| Etc . | | | | |

Version date: 10 December 2020



## ABIVAX ABX464-301 Statistical Analysis Plan

Source: Listing 16.4.5.2

Path\Filename

This layout also applies to:
Table 14.2.4.6.2 Summary of FACIT-Fatigue Score (Efficacy Set 2)



Table 14.2.5.1 Summary of Patients Achieving Different Responses and Remissions (Efficacy Set 1)

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| ARC20 Response | | | | |
| Week 2 | N | xx | xx | xx |
| | Rate | xx.x % | xx.x % | xx.x % |
| | Stratified 95% CI | xx.x % - xx.x % | xx.x % - xx.x % | xx.x % - xx.x % |
| Week 4 | N | xx | XX | XX |
| | Rate | xx.x % | xx.x % | xx.x % |
| | Stratified 95% CI | xx.x % - xx.x % | xx.x % - xx.x % | xx.x % - xx.x % |
| Etc | | | | |
| Etc | | | | |

Source: Listing 16.4.5.3

Path\Filename

Page x/y

Programmer's Note: list of variables consists of ACR20/50/70 response, Categorical DAS28-CRP response, LDA, DAS28-ESR remission, ACR/EULAR remission, SDAI remission, CDAI remission.

This layout also applies to:

Table 14.2.5.2 Summary of Patients Achieving Different Responses and Remissions (Efficacy Set 2)



ABX464-301

#### Table 14.3.1.1 Summary of Adverse Events (Safety Set)

ddMMMyyyy

| | ABX-464<br>100mg<br>(N=xx) | | 100mg 50mg | | | Placebo<br>(N=xx) | | Total (N=xx) |
|---|---|---|---|---|---|---|---|---|
| | n | N (%) | n | N (%) | n | N (%) | n | N (%) |
| Any Adverse Event | xx x | (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Any Treatment-Emergent Adverse Event | xx xx | (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Any Serious Adverse Event | xx xx | (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Adverse Event leading to death | xx x | (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |
| Any grade 3 or higher Adverse Event | xx xx | (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) | xx | xx (xx.x%) |

The table presents number of events (n) and number and percentage of patients (N(%)). The denominator for each percentage is the number of patients within the column.

Source: Listing 16.2.7

Path\Filename



ABX464-301 ddMMMyyyy Table 14.3.1.2.1 Analysis of Treatment-Emergent Adverse Events (Safety Set) ABX-464 ABX-464 Placebo 100mg 50mg p-value (N=xx)(N=xx)(N=xx)Any Treatment-Emergent Adverse Event XX XX XXxx (xx.x%) xx (xx.x%)xx (xx.x%)Yes xx (xx.x%) xx (xx.x%) xx (xx.x%) No Chi-squared test x.xxxx

The denominator for each percentage is the number of patients within the column
TEAE rate between treatments is compared using likelihood ratio chi-square test at a two-sided 10% significance level.

Source: Listing 16.2.7

Path\Filename



Table 14.3.1.2.2 Treatment-Emergent Adverse Events, by SOC and PT: Period 1 (Safety Set)

| | | ABX-4<br>100m<br>(N=x) | g | | ABX-46<br>100mg<br>(N=xx) | | | Placeb<br>(N=xx) | | | Total (N | =xx) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | N (%) | duration<br>(days) | n | N (%) | duration<br>(days) | n | N (%) | duration<br>(days) | n | N (%) | duration<br>(days) |
| Any Treatment-Emergent<br>Adverse Event | xx | xx (xx.x% | ) | xx | xx (xx.x%) | | xx | xx (xx.x%) | | xx | xx (xx.x%) | |
| SOC | xx | xx (xx.x% | ) xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx |
| PT | XX | xx (xx.x% | ) xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx |
| PT | XX | xx (xx.x% | ) xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx |
| SOC<br>Etc | xx | xx (xx.x% | ) xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx | xx | xx (xx.x%) | xx.xx |

Etc

The table presents number of events (n) and number and percentage of patients (N(%)). The denominator for each percentage is the number of patients within the column. Duration (days) represents median duration of AEs (from baseline to occurrence).

Source: Listing 16.2.7

Path\Filename



```
This layout also applies to:

Table 14.3.1.2.3 Treatment-Emergent Adverse Events, by SOC and PT: Period 2 (Safety Set)

Table 14.3.1.3.1 Serious Treatment-Emergent Adverse Events, by SOC and PT: Period 1 (Safety Set)

Table 14.3.1.3.2 Serious Treatment-Emergent Adverse Events, by SOC and PT: Period 2 (Safety Set)

Table 14.3.1.4.1 Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation, by SOC and PT: Period 1 (Safety Set)

Table 14.3.1.4.2 Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation, by SOC and PT: Period 2 (Safety Set)

Table 14.3.1.5.1 Treatment-Emergent Adverse Events of Grade 3 or 4 by SOC and PT: Period 1 (Safety Set)

Table 14.3.1.5.2 Treatment-Emergent Adverse Events of Grade 3 or 4 by SOC and PT: Period 2 (Safety Set)
```



## ABIVAX ABX464-301 Statistical Analysis Plan

ddMMMyyyy

ABX464-301

| Table 14.3.2.1 Listing | of Deaths ( | Safety Set) |
|------------------------|-------------|-------------|
|------------------------|-------------|-------------|

| Treatment | Patient number | Date of death | Cause of death |
|-----------|----------------|---------------|-----------------|
| xxxxxx | xxx-xxxx | ddMMMyyyy | xxxxxxxxxxxxxxx |
| xxxxxx | xxx-xxxx | ddMMMyyyy | xxxxxxxxxxxxxxx |
| Etc | | | |

Path\Filename



#### Table 14.3.2.2 Listing of Serious Adverse Events

| Treatment | Centre/<br>Patient<br>number | Adverse<br>Event<br>PT | Onset date | Resolution<br>date /<br>ongoing | Outcome | Relationship<br>to study<br>drug | Action taken<br>with study drug | Other action<br>taken |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | xxxxxxxxx<br>xxxxxxx<br>xxxx | ddMMMyyyy | ddMMMyyyy /<br>ongoing | Resolved/<br>Resolved<br>without<br>sequelae/<br>Etc | Yes/No | None/ Temporary<br>discontinuation/<br>Etc | Concomitant medication (CM no.)/ Procedure (PR no.) |
| | | xxxxxxxx<br>xxxxxxx<br>xxxx | ddMMMyyyy | ddMMMyyyy /<br>ongoing | Resolved/<br>Resolved<br>without<br>sequelae/<br>Etc | Yes/No | None/ Temporary<br>discontinuation/<br>Etc | Concomitant medication (CM no.)/ Procedure (PR no.) |
| | | Etc | | | | | | |
| Etc | | | | | | | | |
| ath\Filename | | | | | | | | Page x/y |

Version date: 10 December 2020





This layout also applies to: Table 14.3.2.3 Listing of Withdrawals Due to Adverse Events (Safety Set)



ABX464-301

Table 14.3.3.1 Summary of Laboratory Parameters: Haematology (Safety Set)

ABX 464

ABX 464

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|
| aematocrit | | | | | |
| Baseline | N | xx | xx | xx | xx |
| | Mean | xx.xx | xx.xx | xx.xx | xx.xx |
| | SD | XX.XX | XX.XX | xx.xx | xx.xx |
| | SEM | XX.XX | XX.XX | XX.XX | xx.xx |
| | Median | XX.XX | XX.XX | xx.xx | xx.xx |
| | Minimum | XX.X | XX.X | XX.X | xx.x |
| | Maximum | xx.x | xx.x | xx.x | xx.x |
| Week 1 | N | xx | Xx | Xx | Xx |
| | Mean | XX.XX | XX.XX | xx.xx | xx.xx |
| | Etc | | | | |
| Change from baseline to Week 1 | N | xx | Xx | Xx | Xx |
| | Mean | XX.XX | XX.XX | XX.XX | xx.xx |
| | Etc | | | | |
| Etc | | | | | |
| tc | | | | | |

Source: Listing 16.2.8.1



## ABIVAX ABX464-301 Statistical Analysis Plan

Path\Filename

Page x/y

Programming note: start each parameter on a new page

This layout also applies to:

Table 14.3.3.2 Summary of Laboratory Parameters: Biochemistry (Safety Set)



## ABIVAX ABX464-301 Statistical Analysis Plan

ABX464-301 ddMMMyyyy

| Table 14.3.3.3 Listing of Abnormal Laboratory Values (Safet |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

| Treatment | Patient number | Visit | Laboratory Parameter | Value |
|-----------|----------------|--------|----------------------|-------|
| XXXXXX | XXX-XXXX | Week x | xxxxxxxxxxxxxxxx | XX.XX |
| | | | xxxxxxxxxxxxxxx | XX.XX |
| | | | Etc | |
| | | Etc | | |
| | Etc | | | |
| Etc | | | | |

Path\Filename



ABX464-301 ddMMMyyyy

Table 14.3.4 Vital Signs (Safety Set)

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|
| Systolic BP (mmHg) | | | | | |
| Baseline | N | XX | xx | xx | xx |
| | Normal | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal NCS | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal CS | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Mean | xx.xx | xx.xx | xx.xx | xx.xx |
| | SD | xx.xx | XX.XX | xx.xx | XX.XX |
| | SEM | xx.xx | XX.XX | xx.xx | XX.XX |
| | Median | xx.xx | XX.XX | xx.xx | xx.xx |
| | Minimum | xx.x | XX.X | xx.x | xx.x |
| | Maximum | xx.x | XX.X | xx.x | xx.x |
| Week 1 | N | xx | xx | xx | xx |
| | Normal<br>Etc | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Etc | | | | | |
| Etc | | | | | |

The denominator for each percentage is the number of non-missing observations within the column. NCS = Not Clinically Significant; CS = Clinically Significant





Source: Listing 16.4.9

Path\Filename

Page x/y

Programmer's Note: list of variables consists of body temperature, weight, systolic and diastolic blood pressure, heart rate and respiratory rate.



ABX464-301

Table 14.3.5 Shift Table of Physical Examination (Safety Set)

ddMMMyyyy

| | | ABX-464<br>100mg<br>(N=xx) | | ABX-464<br>50mg<br>(N=xx) | | Placebo<br>(N=xx) | | Total<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|
| | | normal | abnormal | normal | abnormal | normal | abnormal | normal | abnormal |
| Eyes | | | | | | | | | |
| Baseline | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Week 1 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Etc | | | | | | | | | |
| Ears | | | | | | | | | |
| Baseline | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Week 1 | N | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Etc | | | | | | | | | |
| Etc | | | | | | | | | |

The denominator for each percentage is the number of non-missing observations within the column.





Source: Listing 16.4.10

Path\Filename

Page x/y

Programmer's Note: list of variables consists of eyes, ears, nose, throat, lungs/thorax, heart/cardiovascular system, abdomen, skin and mucosae, nervous system, lymph nodes, musculo-skeletal system, and, if applicable, others.



ABX464-301

Table 14.3.6 Electrocardiogram (Safety Set)

ddMMMyyyy

| | | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|
| PR interval | | | | | |
| Baseline | N | XX | xx | xx | xx |
| | Normal | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal NCS | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal CS | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Mean | xx.xx | xx.xx | xx.xx | xx.xx |
| | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | xx.xx | xx.xx | xx.xx | xx.xx |
| | Minimum | xx.x | xx.x | xx.x | xx.x |
| | Maximum | xx.x | xx.x | xx.x | xx.x |
| Week 1 | N | xx | xx | xx | xx |
| | Normal<br>Etc | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Etc | | | | | |

Etc

Etc

The denominator for each percentage is the number of non-missing observations within the column. NCS = Not Clinically Significant; CS = Clinically Significant

Source: Listing 16.4.11

Path\Filename





Programmer's Note: The absolute values of PR, QRS, QT and QTc will be summarised at each visit.

XX

xx.xx



Number of dose intakes

Ν

Mean

ABX464-301 ddMMMyyyy

| ADA404-301 | Table 14.3.7 Study Drug Expos | ure and Compliance (Fu | ll Analysis Set) | uunininyyyy |
|---|---|---|---|---|
| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |

XX

XX.XX

XX

XX.XX

| | Mean | xx.xx | xx.xx | xx.xx | xx.xx |
|----------------------------|---------|-------|-------|-------|-------|
| | SD | xx.xx | xx.xx | xx.xx | xx.xx |
| | Median | xx.xx | xx.xx | xx.xx | xx.xx |
| | Minimum | xx.x | xx.x | xx.x | xx.x |
| | Maximum | xx.x | xx.x | xx.x | xx.x |
| Study drug exposure (days) | N | XX | xx | XX | xx |

| | ELC | | | | |
|------------|-----|------------|------------|------------|------------|
| Compliance | N | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Study drug exposure (days) is calculated as (date of last dose) - (date of first dose) + 1.

XX

xx.xx

Source: Listing 16.2.5

Path\Filename Page x/y


Table 14.3.8 Prior Medications (Full Analysis Set)

ddMMMyyyy

| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Any prior medication <sup>1</sup> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X, xxxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XON, xxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X0NXX, xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X0NXX, xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XON, xxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XONXX, xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Etc

WHO-DDE version <XX.X>

The denominator for each percentage is the number of patients in the full analysis set within the column.

Source: Listing 16.4.12.1

<sup>&</sup>lt;sup>1</sup> Medication that stopped prior to date of first dose.



Path\Filename

This layout also applies to: Table 14.3.9.1 Concomitant Medications (Full Analysis Set)



Table 14.3.9.2 Change in Concomitant Medications (Full Analysis Set)

ddMMMyyyy

| | ABX-464<br>100mg<br>(N=xx) | ABX-464<br>50mg<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Any concomitant medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X, xxxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XON, xxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X0NXX, xxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X0NXX, xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XXXXXXXXXXX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XON, xxxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| X0NXX, xxxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| xxxxxxxxxx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Etc | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Etc

WHO-DDE version <XX.X>

The denominator for each percentage is the number of patients in the full analysis set within the column.

Source: Listing 16.4.12.3

Path\Filename







| Listing 16.2 | 2.1.1 | Patient | Disposition |
|--------------|-------|---------|-------------|
|--------------|-------|---------|-------------|

| Treatment | Centre/<br>Patient<br>number | First<br>dose date | Last dose<br>date | Completed<br>study | Date of completion/withdrawal | If not completed specify | Did subject complete the follow-up visit? | Death Date |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-<br>xxxx | ddMMMyyyy | ddMMMyyyy | Yes/No | ddMMMyyyy | specify | Yes/No (specify reason) | ddMMMyyyy |
| | XXX-<br>XXXX | ddMMMyyyy | ddMMMyyyy | Yes/No | ddMMMyyyy | specify | Yes/No (specify reason) | ddMMMyyyy |
| | XXX-<br>XXXX | ddMMMyyyy | ddMMMyyyy | Yes/No | ddMMMyyyy | specify | Yes/No (specify reason) | |
| | XXX-<br>XXXX | ddMMMyyyy | ddMMMyyyy | Yes/No | ddMMMyyyy | specify | Yes/No (specify reason) | |
| Etc | xxx- | ddMMMyyyy | ddMMMyyyy | Yes/No | ddMMMyyyy | specify | Yes/No´(specify | |

Path\Filename



| Listing | 16.2.1.2 | Discontinued | Patients |
|---------|----------|--------------|----------|
|---------|----------|--------------|----------|

| reatment | Centre/<br>Patient number | First dose date | Last dose date | Date of withdrawal | Main reason for withdrawal |
|---|---|---|---|---|---|
| (XXXXX | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ******** |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xxxxxxxxxxxxxxxxxxxxxxxx |

Path\Filename



ABX464-301 ddMMMyyyy

| | Listing 16.2.2 Protocol Deviations | | |
|---|---|---|---|
| Treatment | Centre/<br>Patient<br>number | Major<br>deviation | Protocol deviation |

| XXXXXX | XXX-XXXX | Yes/No | *************************************** |
|--------|----------|--------|-----------------------------------------|
| | xxx-xxxx | Yes/No | |
| | xxx-xxxx | Yes/No | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Etc

XXX-XXXX

Yes/No

Path\Filename



ABX464-301 ddMMMyyyy
Listing 16.2.3 Analysis Datasets

| Treatment | Centre/ Patient number | Full Analysis Set | Per Protocol Set | Safety Set | Efficacy Set 1 | Efficacy Set 2 |
|---|---|---|---|---|---|---|
| www. | VVV VVVV | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| xxxxx | xxx-xxxx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | xxx-xxxx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | xxx-xxxx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Etc | | | | | | |

Path\Filename



| Listing | 16.2.4 | Demographic | Data |
|---------|--------|-------------|------|
|---------|--------|-------------|------|

| Treatment | Centre/<br>Patient<br>number | Date of<br>screening | Date of<br>birth | Age<br>(years) | Gender | Race | Weight<br>(kg) | Height<br>(cm) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | xx | xxxx | xxxx | xx.x | xxx.x | xx.x |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | xx | XXXX | xxxx | xx.x | xxx.x | xx.x |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | xx | XXXX | xxxx | xx.x | xxx.x | xx.x |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | xx | xxxx | xxxx | xx.x | xxx.x | xx.x |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | xx | xxxx | xxxx | xx.x | xxx.x | xx.x |

Etc

Path\Filename



| listing | 16.2.5 | Studv | Drug | Exposure | and | Compliance |
|---------|--------|-------|------|----------|-----|------------|

| Treatment | Centre/<br>Patient<br>number | Date of<br>compliance<br>check | Date of<br>first dose | Date of<br>last dose | Duration of exposure (days) | Capsules<br>used | Capsules<br>expected to be<br>used | Capsules<br>returned | Capsules lost |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | XX | xx | XX |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | xx | xx | xx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | xx | xx | xx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | xx | XX | xx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | xx | XX | xx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | XX | xx | xx | xx |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | xx | xx | xx | XX | xx |
| | Etc | | | | | | | | |

Etc

\*Outside the visit window

Path\Filename



| Listing 16.2.6 | Efficacy | Response | Data: | ACR20/50/70 | Response |
|----------------|----------|----------|-------|-------------|----------|
|----------------|----------|----------|-------|-------------|----------|

| Treatment | Centre/ Patient number | ACR20 Response | ACR50 Response | ACR70 Response |
|---|---|---|---|---|
| xxxxxx | xxx-xxxx | Yes/No | Yes/No | Yes/No |
| | xxx-xxxx | Yes/No | Yes/No | Yes/No |
| | xxx-xxxx | Yes/No | Yes/No | Yes/No |
| | xxx-xxxx | Yes/No | Yes/No | Yes/No |
| Etc | | | | |

Path\Filename



ABX464-301 ddMMMyyyy

Listing 16.2.7 Adverse Event Listing

| Treatment | Centre/<br>Patient<br>number | Baseline<br>date | Adverse<br>Event<br>SOC<br>PT | Onset<br>date | Resolution<br>date<br>/ongoing | Outcome | Serious | Severity | Relationship<br>to study<br>drug | Action taken<br>with study drug | Other<br>action<br>taken |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx-<br>xxxx | ddMMMyyyy | xxxxxxxx<br>xxxxxxx<br>xxxxxxx | ddMMMyyyy | ddMMMyyyy/<br>Ongoing | Resolved/resolved<br>without sequelae<br>/Etc | Yes /No | Grade 1/<br>Grade 2/<br>etc | Yes/No | None /Temporary<br>discontinuation<br>/Etc | Concomitant medication (CM no.)/ Procedure (PR No.) |
| Etc | | ddMMMyyyy | xxxxxxxx<br>xxxxxxx<br>xxxxxxx<br>Etc | ddMMMyyyy | ddMMMyyyy/<br>Ongoing | Resolved/resolved<br>without sequelae<br>/Etc | Yes /No | Grade 1/<br>Grade 2/<br>etc | Yes/No | None /Temporary<br>discontinuation<br>/Etc | Concomitant medication (CM no.)/ Procedure (PR No.) |

Path\Filename



ddMMMyyyy
Listing 16.2.8.1 Laboratory Measurements: Haematology

| Parameter | Treatment | Centre/<br>Patient<br>number | Visit | Was sample taken? | Result | Unit | Investigator's interpretation |
|---|---|---|---|---|---|---|---|
| Haemoglobin | xxxxxxx | xxx-xxxx | Screening | Yes/ No (reason) | xxx.xx | xxxx | Normal/ Abnormal CS/ Abnormal NC |
| | | | Baseline | Yes/ No (reason) | xxx.xx | xxxx | Normal/ Abnormal CS/ Abnormal NC |
| | | | Week 1* | Yes/ No (reason) | xxx.xx | xxxx | Normal/ Abnormal CS/ Abnormal NC |
| | | | Etc | | xxx.xx | xxxx | Normal/ Abnormal CS/ Abnormal NC |
| | | xxx-xxxx | Screening | | xxx.xx | xxxx | Normal/ Abnormal CS/ Abnormal NC |
| | | | Etc | | | | |
| | | Etc | | | | | |
| | Etc | | | | | | |

Etc

\*Outside the visit window CS=Clinically Significant; NCS=Non Clinically Significant

Path\Filename





This layout also applies to:

Listing 16.2.8.2 Laboratory Measurements: Biochemistry

Version date: 10 December 2020



| Listing | 16.4.1 | Final | Status |
|---------|--------|-------|--------|
|---------|--------|-------|--------|

| Treatment | Centre/<br>Patient<br>number | First<br>dose date | Last dose<br>date | Completed<br>treatment | Primary reason for discontinuation (specify) | Was the randomisation code broken? (date and reason) | Will subject enter follow-<br>up? |
|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | Yes/No | xxxxxxxxx<br>(specify) | Yes (ddMMMyyy; xxxxxx)/ No | Yes/No |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | Yes/No | xxxxxxxxx<br>(specify) | Yes (ddMMMyyy; xxxxxx)/ No | Yes/No |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | Yes/No | xxxxxxxxxx<br>(specify) | Yes (ddMMMyyy; xxxxxx)/ No | Yes/No |
| | xxx-xxxx | ddMMMyyyy | ddMMMyyyy | Yes/No | xxxxxxxxx<br>(specify) | Yes (ddMMMyyy; xxxxxx)/ No | Yes/No |
| Etc | | | | | | | |

Path\Filename



ABX464-301 ddMMMyyyy

| Treatment | Centre/ Patient number | Visit | Date |
|-----------|------------------------|-------|-----------|
| XXXXXX | xxx-xxxx | XX | ddMMMyyyy |
| | | xx | ddMMMyyyy |
| | | xx* | ddMMMyyyy |
| | | xx | ddMMMyyyy |
| Etc | | | |

\*Outside the visit window

Path\Filename

ABX464-301 ddMMMyyyy
Listing 16.4.3.1 Inclusion Criteria

| Dnotocol | voncion. | VVVV |
|-----------------|----------|------|
| <b>brofocot</b> | version: | *** |

| Definition of cri | terion |
|-------------------|----------------|
| 1 | xxxxxxxxxxxxxx |
| 2 | xxxxxxxxxxxxxx |
| 3 | Etc |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | |
| Etc | |

Path\Filename

Page x/y

Programmer's Note: The list of criteria will be presented on the first page of the listing. Patient data will start on page 2. Repeat for each protocol amendment if the criteria change.



#### Listing 16.4.3.1 Inclusion Criteria

ddMMMyyyy

| Treatment | Centre/ | Protocol | | | | | Criteria | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient<br>number | version | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Etc |
| xxxxx | xxx-<br>xxxx | x.xx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | xxx-<br>xxxx | x.xx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | xxx-<br>xxxx | x.xx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | xxx-<br>xxxx | x.xx | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

Etc

Path\Filename

Page x/y

This layout also applies to:

Listing 16.4.3.2 Exclusion Criteria



ABX464-301 ddMMMyyyy

#### Listing 16.4.4 Medical History

| Treatment | Centre/<br>Patient number | Date of UC<br>Diagnosis | Any other conditions? | Condition<br>SOC<br>PT | Date of diagnosis | Ongoing/ End date |
|---|---|---|---|---|---|---|
| xxxxxx | xxx-xxxx | ddMMMyyyy | Yes/No | xxxxxxxxxxxx<br>xxxxxxxxxxx<br>xxxxxxxxxx | ddMMMyyyy | Yes/ No<br>(ddMMMyyyy) |
| | | ddMMMyyyy | Yes/No | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ddMMMyyyy | Yes/ No<br>(ddMMMyyyy) |
| Etc | | | | | | |

Path\Filename



Listing 16.4.5.1 Raw Efficacy Data: Individual Components of the ACR20 Response

| Treatment | Centre/<br>Patient<br>number | Visit | C-Reactive<br>Protein<br>(CRP) (mg/L) | Tender/ painful joint count (TJC) (28 joints) | Swollen<br>joint count<br>(SJC) (28<br>joints) | Patient<br>assessment<br>of joint<br>pain (Pain-<br>VAS) | Patient<br>global<br>assessment<br>of disease<br>(PtGA) | Physician's<br>Global<br>Assessment<br>of Disease<br>(PrGA) | HAQ-DI |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx-xxxx | Baseline<br>Etc* | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Etc | | | | | | | | | |

\*Outside the visit window

Path\Filename





ddMMMyyyy

Listing 16.4.5.2 Raw Efficacy Data: ESR, DAS28-CRP, DAS28-ESR, SDAI Score, CDAI Score and FACIT-Fatigue Score

| Treatment | Centre/<br>Patient<br>number | Visit | ESR | DAS28-CRP | DAS28-ESR | SDAI Score | CDAI Score | FACIT-Fatigue Score |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | Baseline<br>Etc* | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |

Etc

\*Outside the visit window

Path\Filename



ABX464-301 ddMMMyyyy

Listing 16.4.5.3 Raw Efficacy Data: Different Responses and Remissions

| Treatment | Centre/<br>Patient<br>number | Visit | Categorical<br>DAS28-CRP<br>response | LDA | DAS28-ESR<br>remission | ACR/EULAR<br>remission | SDAI remission | CDAI remission |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | Baseline<br>Etc* | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| Etc | | | | | | | | |

\*Outside the visit window

Path\Filename



Listing 16.4.9 Vital Signs

| Treatment | Centre/<br>Patient<br>number | Visit | Date of<br>visit | Body<br>temperature<br>(°C) | Weight<br>(kg) | Systolic BP<br>(mmHg) | Diastolic BP<br>(mmHg) | Heart rate<br>(beats/min) | Respiratory<br>rate (/min) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx-xxxx | xx | ddMMMyyyy | xx.x | xx.x | xxx | xxx | xxx | xx.x |
| | | xx | ddMMMyyyy | xx.x | xx.x | xxx | xxx | xxx | xx.x |
| | | xx* | ddMMMyyyy | xx.x | xx.x | xxx | xxx | xxx | xx.x |
| | | XX | ddMMMyyyy | xx.x | XX.X | xxx | xxx | xxx | xx.x |

Etc

Path\Filename

<sup>\*</sup>Outside the visit window



ABX464-301 ddMMMyyyy

| Listing | 16.4.10 | Physical | Examination |
|---------|---------|----------|-------------|
|---------|---------|----------|-------------|

| Treatment | Centre/<br>Patient<br>number | Visit | Date of<br>Visit | Body system | Status | Abnormality |
|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | Screening | ddMMMyyyy | Eyes | Normal/ Abnormal NCS/<br>Abnormal CS/ Not done | ****** |
| | | | | Ear/Nose/Throat | Normal/ Abnormal NCS/<br>Abnormal CS/ Not done | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lungs/Thorax | Normal/ Abnormal NCS/<br>Abnormal CS/ Not done | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Etc | | |
| | | xx* | ddMMMyyyy | Eyes | Normal/ Abnormal NCS/<br>Abnormal CS/ Not done | xxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Etc | | |
| Etc | | | | | | |

\*Outside the visit window

CS=Clinically Significant; NCS=Non Clinically Significant

Path\Filename



#### Listing 16.4.11 12-Lead Electrocardiogram

| Treatment | Centre/<br>Patient<br>number | Visit | Date of<br>visit | Time | PR interval<br>(msec) | QRS width<br>(msec) | QT interval<br>(msec) | QTc interval<br>(msec) | Investigator's interpretation | Abnormality |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXX-<br>XXXX | Baseline | ddMMMyyyy | hh:mm | xx | xx | xx | xx | Normal/<br>Abnormal NCS/<br>Abnormal CS | xxxxxxxxxx |
| | | Week 8 | ddMMMyyyy | hh:mm | xx | xx | XX | xx | Normal/<br>Abnormal NCS/<br>Abnormal CS | xxxxxxxxxx |
| | | Etc* | | | | | | | | |

Etc

Etc

\*Outside the visit window

CS=Clinically Significant; NCS=Non Clinically Significant

Path\Filename



Listing 16.4.12.1 Prior Medications

ddMMMyyyy

| Treatment | Centre/<br>Patient<br>number | Therapy<br>ATC Code<br>PT | Indication | Dose | Unit | Frequency | Route | Start date<br>(Stop date /<br>Ongoing) | Given for pre-<br>existing<br>condition<br>(Related medical<br>history number) | Given for<br>adverse event?<br>(Related adverse<br>event number) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx-xxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxx | xx.x | xxx | xxx | xxx | ddMMMyyyy<br>(ddMMMyyyy) | Yes (xxx) / No | Yes (xxx) / No |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxx | xx.x | xxx | xxx | xxx | ddMMMyyyy<br>(ddMMMyyyy) | Yes (xxx) / No | Yes (xxx) / No |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxx | xx.x | xxx | xxx | xxx | ddMMMyyyy<br>(ddMMMyyyy) | Yes (xxx) / No | Yes (xxx) / No |
| Etc | | | | | | | | | | |

Path\Filename

Page x/y

This layout also applies to:

Listing 16.4.12.2 Concomitant Medications (Programming note: can have stop date as 'ongoing')

Listing 16.4.12.3 Changes to Medications



ABX464-301 ddMMMyyyy

| listing | 16.4.13 | Pregnancy | Test |
|---------|--------------|---------------|------|
| LIJCING | TO . T . T . | i i egilalicy | 1030 |

| Treatment | Centre/<br>Patient number | Visit | Test done | Reason not done | Date of test | Result |
|---|---|---|---|---|---|---|
| xxxxxx | xxx-xxxx | Screening | Yes/No/Not<br>applicable | xxxxxxxxxxx | ddMMMyyyy | Positive/Negative |
| | | xx | Yes/No/Not<br>applicable | xxxxxxxxxxx | ddMMMyyyy | Positive/Negative |
| | | xx* | Yes/No/Not<br>applicable | xxxxxxxxxxx | ddMMMyyyy | Positive/Negative |
| | | xx | Yes/No/Not<br>applicable | xxxxxxxxxxx | ddMMMyyyy | Positive/Negative |
| | | Etc | | | | |

Etc

\*Outside the visit window

Path\Filename



| Listing | 16.4.14 | Laboratory | Samples | Collection |
|---------|---------|------------|---------|------------|
|---------|---------|------------|---------|------------|

| Parameter xxxxxx | Treatment<br>xxxxxx | Centre/<br>Patient<br>number | Visit<br>Screening | Sample<br>taken<br>Yes/No | Reason not<br>done | Date of<br>test | Result | Interpretation |
|---|---|---|---|---|---|---|---|---|
| | | | | | xxxxxxxxxxx | ddMMMyyyy | xx | Normal/ Abnormal CS/ Abnormal NCS |
| | | | xx | Yes/No | xxxxxxxxxxx | ddMMMyyyy | XX | Normal/ Abnormal CS/ Abnormal NCS |
| | | | xx* | Yes/No | xxxxxxxxxxx | ddMMMyyyy | xx | Normal/ Abnormal CS/ Abnormal NCS |
| | | | XX | Yes/No | xxxxxxxxxxx | ddMMMyyyy | xx | Normal/ Abnormal CS/ Abnormal NCS |
| | | | Etc | | | | | |

Etc

\*Outside the visit window

CS=Clinically Significant; NCS=Non Clinically Significant

Path\Filename

Page x/y

Version date: 10 December 2020



### 16 APPENDICES

#### 16.1 STUDY FLOWCHART

| | Screening<br>Period | | Study Treatment Period | | | | | Follow-<br>up<br>Period |
|---|---|---|---|---|---|---|---|---|
| | D-30 to D-I | D0 | D7 | DI4 | D28 | D56 | D84 | D105 |
| | | W0 | WI | W2 | W4 | W8 | WI2 | WI5 |
| Time Window (time between two visits≤30 days) | | | ± 2 days | ± 2<br>days | ± 2 days | ± 2 days | ± 2 days | ± 2 days |
| | Screening | <b>Baseline</b> | VI | V2 | V3 | V4 | V5 | EOS |
| Obtained Inform Consent | Х | | | | | | | |
| Check of IN/EX Criteria | Х | | | | | | | |
| Medical History | Х | | | | | | | |
| Height Measurement (cm) | Х | | | | | | | |
| Body Weight (kg) | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical Examination | X | X | X | X | X | X | X | X |
| Vital signs | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X |
| ECG (12 lead) | X | X | ^ | | | _^_ | X | X* |
| Blood Pregnancy test (WOCBP) | X | | | | X | Х | X | X |
| Urine Pregnancy test (WOCBP) | <del> ^</del> | Х | | | | _^ | _^ | _^_ |
| | - | | | | | | | |
| Randomization | - | X | | | | | | |
| ABX464/placebo treatment dispensation | | X | | | X | X | | |
| Hematology + Biochemistry# | X# | Х | Х | X | Х | X | Х | X |
| Blood samples drug PK (pre-dose) | | | | Х | | Х | | X** |
| Blood samples drug PK | | X | | Х | | X | | |
| (I-, 2- & 3- hours post-dose) | | | | | | | | |
| Blood samples for Cytokines (gel tube) | | Х | Х | X | X | Х | Х | |
| <b>Blood samples for Cytokines (</b> Truculture® tube <b>)</b> | | Х | | | | X | | |
| Blood samples for flow cytometry cells count*** | | X | | | | × | | |
| Blood samples for CRP, ESR | Х | Х | X | Х | Х | Х | Х | |
| Blood samples for miR-124 (Paxgene® | _ ^ | | | | | | | |
| tube) | | × | | | | Х | | |
| Tender Joint Count (28) | Х | Х | | Х | Х | Х | Х | |
| Swollen Joint Count (28) | X | Х | | X | Х | Х | Х | |
| Patient Global Assessment of Disease (PtGA-VAS) | Х | Х | | Х | X | Х | Х | |
| Patient assessment of Joint Pain (Pain-VAS) | | X | | X | Х | Х | X | |
| Investigator Global Assessment of Disease (PrGA-VAS) | | X | | Х | X | Х | X | |
| Health Assessment Questionnaire - Disease Index (HAQ-DI) | | Х | | Х | Х | × | Х | |
| Functional Assessment of Chronic Illness<br>Therapy (FACIT)-Fatigue | | Х | | Х | X | X | Х | |
| Patient diary (dispensation/check) | | Х | Х | Х | Х | Х | Х | |
| Adverse Events recording | X | X | X | X | X | X | X | Х |
| Follow_up Headache Questionnaire in case of persistent headache (see section 5.3.2) | | X (throughout the study, if needed) | | | | | | |
| Dermatologist consultation in case of skin effect (see section 5.3.2) | *566 | X (throughout the study, if needed) FOS visit in case of early termination only: **trough levels PK samples: | | | | | | |

<sup>#</sup>Tests of TB, HIV, HCV, HBV only at screening; \*ECG at EOS visit in case of early termination only; \*\*trough levels PK samples; \*\*\*Only in French Coordinating Investigator's Site; Two visits should not be conducted more than 30 days apart